

# A PHASE 3, RANDOMIZED, OBSERVER-BLIND STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF MULTIPLE FORMULATIONS OF THE VACCINE CANDIDATE BNT162b2 AGAINST COVID-19 IN HEALTHY ADULTS 18 THROUGH 55 YEARS OF AGE

Study Sponsor: BioNTech

**Study Conducted By:** Pfizer

**Study Intervention Number:** PF-07302048

**Study Intervention Name:** BNT162b2 RNA-Based COVID-19 Vaccine

US IND Number: 19736

**EudraCT Number:** 2020-002641-42 **ClinicalTrials.gov ID:** NCT04816669

**Protocol Number:** C4591020

Phase: 3

**Short Title:** A Phase 3 Study to Evaluate the Safety, Tolerability, and Immunogenicity of Multiple Formulations of BNT162b2 Against COVID-19 in Healthy Adults

This document and accompanying materials contain confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing these documents, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

# **Protocol Amendment Summary of Changes Table**

| <b>Document History</b> | | |
|---|---|---|
| Document | Version Date | Summary and Rationale for Changes |
| Protocol amendment 2 | 13 Sep 2021 | <ul> <li>The primary immunogenicity analysis demonstrated that the immune response elicited by the lyophilized formulation did not meet the noninferiority criteria compared to the frozen-liquid formulation of BNT162b2. As a result, for the benefit of participants, updates were made to offer and administer an additional vaccine dose, using the frozen-liquid formulation, to participants who originally received 2 doses of the lyophilized formulation of BNT162b2.</li> <li>Exploratory estimand relating to lyophilized formulation have been reported (GMRs of RTU formulation to lyophilized formulation in SDVs 1 month after Dose 2)</li> <li>Added 2 exploratory objectives corresponding to administration of Dose 3 and updated the pertinent details for the statistical analysis.</li> <li>Updated Section 9.4.4 to add an exploratory immunogenicity objective, and clarified that IgG data from all participants in Part 1 will be used and neutralizing titer data from a random sample of ~30 age-matched participants in Part 1 receiving frozen-liquid BNT162b2 in MDVs will be used.</li> <li>Following updates were in specified sections in response to commitment made to CBER concerning myocarditis and pericarditis: <ul> <li>Updated Section 2.3.1</li> <li>(Risk Assessment) to address myocarditis and pericarditis safety concerns.</li> <li>Added Section 8.13 for requirement of unplanned visit to capture data pertaining to myocarditis and pericarditis.</li> </ul> </li> </ul> |

| Protocol amendment 1 Original protocol | 15 Apr 2021 | <ul> <li>Removed all references to lyophilized MDV and added ability to assess frozen-liquid BNT162b2 with LNP size at the upper end of specification and RTU BNT162b2 in a second part of the study.</li> <li>Updated corresponding objectives, estimands, and endpoints, including removal of 1 Primary Immunogenicity objective and addition of 2 new Exploratory objectives in line with changes to formulation evaluation. Section 9 (Statistical Considerations) was updated in line with the changes to objectives, estimands, and endpoints.</li> <li>Updated the planned number of participants required for Part 2 of the study.</li> <li>Removed review of temporary delay of vaccination criteria at Visit 1 in SoA and Section 8.11.1 (Visit 1) and revised text in Section 5.5 (Temporary Delay Criteria).</li> <li>Updated Section 2.3.1.</li> <li>Addressed discrepancy in Section 8.11.1 (Visit 1) describing site staff responsibilities for the IRT system entries (Impala) compared with text in the Impala quick reference guide, IP manual, and site blinding plan.</li> <li>Updated Section 10.4.1 (Male Participant Reproductive Inclusion Criteria) to correct a typographical error.</li> </ul> |
|---|---|---|
| C 1 | | |

This amendment incorporates all revisions to date, including amendments made at the request of country health authorities and IRBs/ECs.

# **TABLE OF CONTENTS**

| LIST OF TABLES | 8 |
|---|---|
| 1. PROTOCOL SUMMARY | 9 |
| 1.1. Synopsis | 9 |
| 1.2. Schema | 13 |
| 1.3. Schedule of Activities | 14 |
| 1.3.1. Schedule of Activities for Those Participants Who Originally Received Lyophilized Formulation and Accept the Offer to Receive Current Frozen Formulation of BNT162b2 | 16 |
| 2. INTRODUCTION | 18 |
| 2.1. Study Rationale | 18 |
| 2.2. Background | 18 |
| 2.2.1. Clinical Overview | 19 |
| 2.3. Benefit/Risk Assessment | 22 |
| 2.3.1. Risk Assessment | 24 |
| 2.3.2. Benefit Assessment | 26 |
| 2.3.3. Overall Benefit/Risk Conclusion | 26 |
| 3. OBJECTIVES, ESTIMANDS, AND ENDPOINTS | 26 |
| 4. STUDY DESIGN | 27 |
| 4.1. Overall Design | 27 |
| 4.2. Scientific Rationale for Study Design | 28 |
| 4.3. Justification for Dose | 29 |
| 4.4. End of Study Definition | 29 |
| 5. STUDY POPULATION | 29 |
| 5.1. Inclusion Criteria | 29 |
| 5.2. Exclusion Criteria | 30 |
| 5.3. Lifestyle Considerations | 31 |
| 5.3.1. Contraception. | 31 |
| 5.4. Screen Failures | 31 |
| 5.5. Criteria for Temporarily Delaying Enrollment/Randomization/Study Intervention Administration | 32 |
| 6. STUDY INTERVENTION | 33 |
| 6.1. Study Intervention(s) Administered | 33 |

| 6.1.1. Administration | 33 |
|---|---|
| 6.2. Preparation/Handling/Storage/Accountability | 34 |
| 6.2.1. Preparation and Dispensing | 35 |
| 6.3. Measures to Minimize Bias: Randomization and Blinding | 35 |
| 6.3.1. Allocation to Study Intervention | 35 |
| 6.3.2. Blinding of Site Personnel | 36 |
| 6.3.3. Blinding of the Sponsor | 36 |
| 6.3.4. Breaking the Blind | 37 |
| 6.4. Study Intervention Compliance | 37 |
| 6.5. Concomitant Therapy | 37 |
| 6.5.1. Prohibited During the Study | 37 |
| 6.5.2. Permitted During the Study | 38 |
| 6.6. Dose Modification | 38 |
| 6.7. Intervention After the End of the Study | 38 |
| 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL | 39 |
| 7.1. Discontinuation of Study Intervention | 39 |
| 7.2. Participant Discontinuation/Withdrawal From the Study | 39 |
| 7.2.1. Withdrawal of Consent | 40 |
| 7.3. Lost to Follow-up | 40 |
| 8. STUDY ASSESSMENTS AND PROCEDURES | 41 |
| 8.1. Efficacy and/or Immunogenicity Assessments | 42 |
| 8.1.1. Biological Samples | 42 |
| 8.2. Safety Assessments | 43 |
| 8.2.1. Clinical Safety Laboratory Assessments | 43 |
| 8.2.2. Electronic Diary | 43 |
| 8.2.2.1. Grading Scales | 44 |
| 8.2.2.2. Local Reactions | 44 |
| 8.2.2.3. Systemic Events | 45 |
| 8.2.2.4. Fever | 46 |
| 8.2.2.5. Antipyretic Medication | 46 |
| 8.2.3. Pregnancy Testing | 46 |

| 8.3. Adverse Events and Serious Adverse Events | 47 |
|---|---|
| 8.3.1. Time Period and Frequency for Collecting AE and SAE Information | 47 |
| 8.3.1.1. Reporting SAEs to Pfizer Safety | 48 |
| 8.3.1.2. Recording Nonserious AEs and SAEs on the CRF | 48 |
| 8.3.2. Method of Detecting AEs and SAEs | 48 |
| 8.3.3. Follow-up of AEs and SAEs | 48 |
| 8.3.4. Regulatory Reporting Requirements for SAEs | 49 |
| 8.3.5. Exposure During Pregnancy or Breastfeeding, and Occupational Exposure | 49 |
| 8.3.5.1. Exposure During Pregnancy | 49 |
| 8.3.5.2. Exposure During Breastfeeding | 51 |
| 8.3.5.3. Occupational Exposure | 51 |
| 8.3.6. Cardiovascular and Death Events | 51 |
| 8.3.7. Disease-Related Events and/or Disease-Related Outcomes Not Qualifying as AEs or SAEs | 51 |
| 8.3.8. Adverse Events of Special Interest | 52 |
| 8.3.8.1. Lack of Efficacy | 52 |
| 8.3.9. Medical Device Deficiencies | 52 |
| 8.3.10. Medication Errors | 52 |
| 8.4. Treatment of Overdose | 53 |
| 8.5. Pharmacokinetics | 53 |
| 8.6. Pharmacodynamics | 53 |
| 8.7. Genetics | 53 |
| 8.8. Biomarkers | 54 |
| 8.9. Immunogenicity Assessments | 54 |
| 8.10. Health Economics | 54 |
| 8.11. Study Procedures | 54 |
| 8.11.1. Visit 1 – Vaccination 1 (Day 1) | 54 |
| 8.11.2. Visit 2 – Vaccination 2 (19 to 23 Days After Visit 1) | 56 |
| 8.11.3. Visit 3 – 1-Month Follow-up (28 to 35 Days After Visit 2) | 59 |
| 8.11.4. Unscheduled Visits for a Grade 3 or Suspected Grade 4 Reaction | 59 |
| 8.12. Study Procedures for Participants Who Accept the Offer to Receive Dose 3 | 60 |
| 8.12.1. Visit 101 – Vaccination 3 (At Least 90 Days After Visit 2) | 60 |

| 8.12.2. Visit 102 – 1-Month Follow-up (28 to 35 Days After Visit 101) | 63 |
|---|---|
| 8.13. Additional Procedures for Monitoring of Potential Myocarditis or | 62 |
| Pericarditis | |
| 9. STATISTICAL CONSIDERATIONS | |
| 9.1. Estimands and Statistical Hypotheses | |
| 9.1.1. Estimands | |
| 9.1.2. Statistical Hypothesis | |
| 9.1.3. Multiplicity Considerations | |
| 9.2. Sample Size Determination | |
| 9.3. Analysis Sets | |
| 9.4. Statistical Analyses | 66 |
| 9.4.1. General Considerations | 66 |
| 9.4.1.1. Analysis for Binary Data | 67 |
| 9.4.1.2. Analysis for Continuous Data | 67 |
| 9.4.2. Primary Endpoint(s) | 68 |
| 9.4.3. Secondary Endpoint(s) | 68 |
| 9.4.4. Exploratory Endpoint(s) | 69 |
| 9.5. Interim Analyses | 70 |
| 9.6. Data Monitoring Committee or Other Independent Oversight Committee | 70 |
| 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | 71 |
| 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations | 71 |
| 10.1.1. Regulatory and Ethical Considerations | 71 |
| 10.1.1.1. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP | |
| 10.1.2. Financial Disclosure | 72 |
| 10.1.3. Informed Consent Process | 72 |
| 10.1.4. Data Protection | 73 |
| 10.1.5. Dissemination of Clinical Study Data | |
| 10.1.6. Data Quality Assurance | |
| 10.1.7. Source Documents | |
| 10.1.8. Study and Site Start and Closure | |
| 10.1.9. Publication Policy | |
| · | |

| 1 | 0.1.10. Sponsor's Qualified Medical Personnel | 77 |
|---|---|---|
| 10.2. A | ppendix 2: Clinical Laboratory Tests | 78 |
| | ppendix 3: Adverse Events: Definitions and Procedures for Recording, luating, Follow-up, and Reporting | 79 |
| 1 | 0.3.1. Definition of AE | 79 |
| 1 | 0.3.2. Definition of SAE | 80 |
| 1 | 0.3.3. Recording/Reporting and Follow-up of AEs and/or SAEs | 82 |
| 1 | 0.3.4. Reporting of SAEs | 85 |
| 10.4. A | ppendix 4: Contraceptive Guidance | 86 |
| 1 | 0.4.1. Male Participant Reproductive Inclusion Criteria | 86 |
| 1 | 0.4.2. Female Participant Reproductive Inclusion Criteria | 86 |
| 1 | 0.4.3. Woman of Childbearing Potential | 87 |
| 1 | 0.4.4. Contraception Methods | 88 |
| 10.5. A | ppendix 5: Liver Safety: Suggested Actions and Follow-up Assessments | 90 |
| 10.6. A | ppendix 6: Abbreviations | 92 |
| 11. REFERE | NCES | 95 |
| | LIST OF TABLES | |
| Table 1. | Local Reaction Grading Scale | 44 |
| Table 2. | Systemic Event Grading Scale | 45 |
| Table 3. | Scale for Fever | 46 |
| Table 4. | Power Analysis for Noninferiority Assessment | 65 |

#### 1. PROTOCOL SUMMARY

### 1.1. Synopsis

**Short Title:** A Phase 3 Study to Evaluate the Safety, Tolerability, and Immunogenicity of Multiple Formulation of BNT162b2 Against COVID-19 in Healthy Adults

#### Rationale

A pneumonia of unknown cause detected in Wuhan, China, was first reported in December 2019. In January 2020, the pathogen causing this outbreak was identified as a novel coronavirus 2019. The outbreak was declared a Public Health Emergency of International Concern on 30 January 2020. On 12 February 2020, the virus was officially named as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), and the WHO officially named the disease caused by SARS-CoV-2 as coronavirus disease 2019 (COVID-19). On 11 March 2020, the WHO upgraded the status of the COVID-19 outbreak from epidemic to pandemic, which continues to spread globally at high speed.

Based on Phase 2/3 safety, immunogenicity, and efficacy data, BNT162b2 was shown to be effective and has been authorized for temporary or emergency use in multiple countries.

The Pfizer-BioNTech COVID-19 vaccine (also referred to as BNT162b2) is administered intramuscularly as a 2-dose series spaced 21 days apart at a dose of 30 µg each. Study C4591001 (NCT04368728) is an ongoing Phase 1/2/3 trial in ~44,000 participants designed to generate safety, tolerability, immunogenicity, and efficacy data from a novel RNA-based vaccine candidate. The trial is being conducted in a heterogeneous study population: eligible participants  $\geq 12$  years of age, healthy participants, including those participants with stable chronic medical conditions, including HIV-, HCV-, and HBV-positive participants. The study consists of 2 parts: Phase 1: to identify the preferred vaccine candidate (BNT162b1 or BNT162b2) and dose level (10 μg, 20 μg, 30 μg, or 100 μg [for BNT162b1]); Phase 2/3: an expanded-cohort and efficacy part for the selected vaccine candidate (BNT162b2). BNT162b2 was selected from the Phase 1 part of this study based on the overall safety, tolerability, and immunogenicity. Vaccine efficacy from Phase 2/3 for the primary endpoint against confirmed COVID-19 occurring at least 7 days after the second dose was 95% with 8 COVID-19 cases in the active vaccine group compared to 162 COVID-19 cases in the placebo group. Data from approximately 38,000 participants randomized 1:1 with a median of 2 months of follow-up after the second dose of vaccine showed a favorable safety profile at a dose of 30 µg in participants 16 years of age and older.

To optimize storage and distribution of this vaccine on a wide scale, a lyophilized or alternate formulation that will be stable at standard refrigerator or freezer temperatures is required. Therefore, this study will compare the safety and tolerability of lyophilized BNT162b2 presented in SDVs to those of frozen-liquid BNT162b2 in MDVs and determine whether the immune response is noninferior. Separately, the study will also describe the safety and immunogenicity of frozen-liquid BNT162b2 with LNP size at the upper end of specification and RTU BNT162b2 (the immediate manufacturing precursor to the lyophilate).

The primary immunogenicity analysis demonstrated that the immune response elicited by the lyophilized formulation did not meet the noninferiority criteria compared to the frozen-liquid formulation of BNT162b2. As a result, for the benefit of participants, all study participants who received 2 doses of the lyophilized formulation will be offered an additional vaccine dose, using the 30-µg dose of frozen-liquid formulation of BTN162b2.

# Objectives, Estimands, and Endpoints

| Objectives | Estimands | Endpoints |
|---|---|---|
| Primary Immunogenicity | | |
| To demonstrate that the immune response induced by lyophilized BNT162b2 in SDVs is noninferior to the immune response induced by frozen-liquid BNT162b2 in MDVs in participants without evidence of SARS-CoV-2 infection during the study | In participants complying with the key protocol criteria (evaluable participants): • GMR of lyophilized formulation in SDVs to frozen-liquid formulation in MDVs 1 month after Dose 2 | Full-length S-binding IgG levels |
| | Primary Safety | |
| To evaluate the safety of BNT162b2 when administered on a 2-dose schedule in healthy adults 18 through 55 years of age | In participants receiving at least 1 dose of study intervention from each vaccine group, the percentage of participants reporting: • Local reactions for up to 7 days following each dose • Systemic events for up to 7 days following each dose • AEs and SAEs from Dose 1 through 1 month after Dose 2 | <ul> <li>Local reactions (pain at the injection site, redness, and swelling)</li> <li>Systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain)</li> <li>AEs</li> <li>SAEs</li> </ul> |
| | Secondary Immunogenicity | |
| To describe the immune responses induced by lyophilized BNT162b2 in SDVs and frozen-liquid BNT162b2 in MDVs | In evaluable participants from each vaccine group: GMCs at baseline (before Dose 1) and 1 month after Dose 2 GMFR from baseline (before Dose 1) to 1 month after Dose 2 | Full-length S-binding IgG levels |
| Exploratory | | |
| To describe the immune responses induced by frozen-liquid BNT162b2 with LNP size at the upper end of specification and RTU BNT162b2 in participants without evidence of SARS-CoV-2 infection during the study | In evaluable participants: • GMR of frozen-liquid BNT162b2 with LNP size at the upper end of specification to frozen-liquid BNT162b2 in MDVs 1 month after Dose 2 | Full-length S-binding IgG<br>levels and/or SARS-CoV-2<br>neutralizing titers |

| Objectives | Estimands | Endpoints |
|---|---|---|
| To describe the immune responses induced by frozenliquid BNT162b2 with LNP size at the upper end of specification and RTU BNT162b2 | In evaluable participants from each vaccine group: GMCs and/or GMTs at baseline (before Dose 1) and 1 month after Dose 2 GMFR from baseline (before Dose 1) to 1 month after Dose 2 | Full-length S-binding IgG<br>levels and/or SARS-CoV-2<br>neutralizing titers |
| To describe the safety profile of frozen-liquid BNT162b2 formulation when given as a third dose to participants who originally received 2 doses of the lyophilized formulation of BNT162b2 | <ul> <li>In participants who originally received 2-dose series of the lyophilized formulation of BNT162b2:</li> <li>Local reactions for up to 7 days following third dose</li> <li>Systemic events for up to 7 days following third dose</li> <li>AEs from Dose 3 to 1 month after Dose 3</li> <li>SAEs from Dose 3 to 1 month after Dose 3</li> </ul> | <ul> <li>Local reactions (pain at the injection site, redness, and swelling)</li> <li>Systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain)</li> <li>AEs</li> <li>SAEs</li> </ul> |
| To describe the immune response elicited by frozen-liquid BNT162b2 formulation when given as a third dose following a primary series of lyophilized BNT162b2 | In evaluable participants who originally received a 2-dose series of the lyophilized formulation of BNT162b2 GMFR from prior to Dose 3 to 1 month after Dose 3 GMCs and/or GMTs at baseline, at 1 month after Dose 2, prior to Dose 3, and 1 month after Dose 3 | Full-length S-binding IgG<br>levels and/or SARS-CoV-2<br>neutralizing titers |

# **Overall Design**

This is a Phase 3, randomized, observer-blind study to evaluate the safety, tolerability, and immunogenicity of multiple formulations of BNT162b2, an RNA-based COVID-19 vaccine, administered on a 2-dose schedule in healthy adults 18 through 55 years of age. In Part 1, participants will be randomized in a 1:1 ratio to 1 of the 2 groups (lyophilized SDV or frozen-liquid MDV control for lyophilized SDV). Separately, in Part 2, participants will be randomized in a 1:1 ratio to 1 of the 2 groups (frozen-liquid BNT162b2 with LNP size at the upper end of specification or RTU BNT162b2). The duration of the study for each participant will be approximately 2 months. The study will be conducted in the US with potential to expand to other countries.

Updates as part of protocol amendment 2:

All participants who originally received 2 doses of the lyophilized formulation of BNT162b2 will be offered the opportunity to receive a third dose with the current frozen-liquid formulation of BNT162b2. Those participants who accept the offer of receiving a third dose will have 2 additional visits. The study duration will be extended for 1 additional month for those participants who accept the offer of receiving a third dose.

#### **Number of Participants**

Approximately 550 participants will be randomly assigned in a 1:1 ratio to either lyophilized SDV or frozen-liquid MDV control for lyophilized SDV; separately, approximately 60 participants will be randomly assigned in a 1:1 ratio to either frozen-liquid BNT162b2 with LNP size at the upper end of specification or RTU BNT162b2, for a total of approximately 610 randomized participants. It is expected that approximately 488 evaluable participants will complete the study, based on a 20% nonevaluable rate.

#### Data Monitoring Committee or Other Independent Oversight Committee: Yes

This study will use a DMC. The DMC is independent of the study team and includes external members. The DMC charter describes the role of the DMC in more detail.

The DMC will be responsible for ongoing monitoring of the safety of participants in the study according to the charter. This may include, but is not limited to:

- Contemporaneous review of related AEs up to 1 month after completion of the vaccination schedule,
- Contemporaneous review of all SAEs up to 1 month after completion of the vaccination schedule.

The recommendations made by the DMC to alter the conduct of the study will be forwarded to the appropriate Pfizer personnel for final decision. Pfizer will forward such decisions, which may include summaries of aggregate analyses of safety data, to regulatory authorities, as appropriate.

#### **Statistical Methods**

The primary immunogenicity objective will be evaluated by a formal hypothesis test for noninferiority of the full-length S-binding IgG levels induced by lyophilized SDV compared to the corresponding frozen-liquid MDV BNT162b2 control. GMRs will be provided along with associated 2-sided 95% CIs. Noninferiority will be declared if the lower bound of the 2-sided 95% CI for the GMR of lyophilized BNT162b2 relative to frozen-liquid MDV BNT162b2 is greater than 0.67 (using a 1.5-fold noninferiority criterion).

With 220 evaluable participants in each of the 2 vaccine groups in Part 1, the study has a power of 90.1% for declaring noninferiority of lyophilized BNT162b2 to frozen-liquid MDV BNT162b2. Assuming a nonevaluable rate of 20%, the study will randomize approximately 275 participants to each group in Part 1 of the study to achieve the required number of evaluable participants.

The secondary immunogenicity objective will be evaluated descriptively by GMCs, GMFRs, and the associated 95% CIs for the full-length S-binding IgG levels for each vaccine group.

The primary safety objective will be evaluated by descriptive statistics including counts and percentages of participants and the associated Clopper-Pearson 95% CIs for local reactions, systemic events, and AEs/SAEs for each vaccine group.

#### 1.2. Schema

| Randomization<br>Ratio | Randomized | Visit 1<br>Vaccination 1 | | Visit 2<br>Vaccination 2 | | Visit 3<br>1-Month Follow-Up |
|---|---|---|---|---|---|---|
| 1 | 275 | Lyophilized SDV | 21 Days | Lyophilized SDV | 1 Month | Blood Sampling<br>Nasal Swab |
| 1 | 275 | Frozen-liquid MDV<br>(control for lyo SDV) | 21 Days | Frozen-liquid MDV<br>(control for lyo SDV) | 1 Month | Blood Sampling<br>Nasal Swab |
| Fro | • , | LNP size at the upper en<br>cipants will be randomiz | - | , | - | parately |
| 1 | 30 | Frozen-liquid MDV<br>(LNP size at the upper end<br>of specification) | 21 Days | Frozen-liquid MDV<br>(LNP size at the upper end<br>of specification) | 1 Month | Blood Sampling<br>Nasal Swab |
| 1 | 30 | RTU | 21 Days | RTU | 1 Month | Blood Sampling<br>Nasal Swab |
| | | Blood Sampling<br>Nasal Swab | | | | |

Note: As part of protocol amendment 2, all participants who originally received 2 doses of the lyophilized formulation of BNT162b2 will be offered the opportunity to receive a third dose of the frozen-liquid formulation of BNT162b2.

#### 1.3. Schedule of Activities

The SoA table provides an overview of the protocol visits and procedures. Refer to the Study Assessments and Procedures section of the protocol for detailed information on each procedure and assessment required for compliance with the protocol.

The investigator may schedule visits (unplanned visits) in addition to those listed in the SoA table, in order to conduct evaluations or assessments required to protect the well-being of the participant.

| Visit Number | 1 | 2 | 3 |
|---|---|---|---|
| Visit Description | Vaccination 1 | Vaccination 2 | 1-Month Follow-up Visit |
| Visit Window | Day 1 <sup>a</sup> | 19 to 23 Days After Visit 1 | 28 to 35 Days After Visit 2 |
| Obtain informed consent | X | | |
| Assign participant number | X | | |
| Obtain demography and medical history data | X | | |
| Perform clinical assessment <sup>b</sup> | X | | |
| Measure height and weight | X | | |
| Measure temperature (body) | X | X | |
| Perform urine pregnancy test (if appropriate) | X | X | |
| Confirm use of contraceptives (if appropriate) | X | X | X |
| Collect nonstudy vaccine information | X | X | X |
| Collect prohibited medication use | | X | X |
| Confirm eligibility | X | X | |
| Review temporary delay criteria | | X | |
| Collect blood sample for immunogenicity assessment & for serological testing for prior COVID-19 infection <sup>c</sup> | ~20 mL | | ~20 mL |
| Obtain nasal (midturbinate) swab for determination of current SARS-CoV-2 status <sup>c</sup> | X | | X |
| Obtain randomization number and study intervention allocation | X | | |
| Administer study intervention | X | X | |

| Visit Number | 1 | 2 | 3 |
|---|---|---|---|
| Visit Description | Vaccination 1 | Vaccination 2 | 1-Month Follow-up Visit |
| Visit Window | Day 1 <sup>a</sup> | 19 to 23 Days After Visit 1 | 28 to 35 Days After Visit 2 |
| Assess acute reactions for at least 30 minutes after study intervention administration | X | X | |
| Explain/review participant communication methods (including for reactogenicity e-diary completion), assist the participant with downloading the app, or issue provisioned device, if required | X | X | |
| Provide/ensure participant has a thermometer and measuring device | X | X | |
| Review reactogenicity e-diary data (daily review is optimal during the active diary period) | $X \rightarrow$ | $X \rightarrow$ | |
| Review ongoing reactogenicity e-diary symptoms with participant and obtain stop dates | | X | X |
| Collect AEs and SAEs | X | X | $X^{d}$ |
| Collect e-diary or assist the participant to delete the application | | | X |

Abbreviations:  $\rightarrow$  = continuous/ongoing event; e-diary = electronic diary.

- a. The visit may be conducted across 2 consecutive days; if so, all steps from assessing the inclusion and exclusion criteria onward must be conducted on the same day.
- b. Including, if indicated, a physical examination.
- c. Administration of study intervention is not dependent on test results.
- d. Any AEs occurring up to 48 hours after blood draw and nasal swab collection must be recorded.

# 1.3.1. Schedule of Activities for Those Participants Who Originally Received Lyophilized Formulation and Accept the Offer to Receive Current Frozen Formulation of BNT162b2

| Visit Number | 101 | 102 |
|---|---|---|
| Visit Description | Vaccination 3 | 1-Month Follow-up Visit 28 to 35 Days After Visit 101 |
| Visit Window | At Least 90 Days After Vaccination 2 | |
| Obtain informed consent | X | |
| Confirm participant originally received BOTH doses of lyophilized formulation of BNT162b2 | X | |
| Measure prevaccination temperature (body) | X | |
| Perform urine pregnancy test (if appropriate) | X | |
| Confirm use of contraceptives (if appropriate) | X | X |
| Collect nonstudy vaccine information | X | X |
| Collect prohibited medication use | X | X |
| Review and consider eligibility <sup>a</sup> | X | |
| Review temporary delay criteria | X | |
| Collect blood sample for immunogenicity assessment | ~20 mL | ~20 mL |
| Obtain nasal (midturbinate) swab for determination of current SARS-CoV-2 status <sup>b</sup> | X | X |
| Obtain study intervention allocation using the IRT system | X | |
| Administer study intervention | X | |
| Assess acute reactions for at least 30 minutes after study intervention administration | X | |
| Provide thermometer and measuring device | X | |
| Remind participant of e-diary technologies | X | |
| Review reactogenicity e-diary data (daily review is optimal during the active diary period) | X | |

| Visit Number | 101 | 102 |
|---|---|---|
| Visit Description | Vaccination 3 | 1-Month Follow-up Visit |
| Visit Window | At Least 90 Days After Vaccination 2 | 28 to 35 Days After Visit 101 |
| Review ongoing reactogenicity e-diary symptoms and obtain stop dates | X | X |
| Collect AEs and SAEs as appropriate <sup>c</sup> | X | X <sup>c</sup> |
| Collect e-diary or assist the participant to delete application | | X |

Abbreviations: e-diary = electronic diary; IRT = interactive response technology.

- a. Confirm that the participant meets all of the inclusion criteria and does not meet exclusion criteria 1, 3, 5, 6, 7, 10, 11, 12, 13, and 14.
- b. Administration of study intervention is not dependent on test results
- c. Any AEs occurring up to 48 hours after blood draw and nasal swab collection must be recorded.

#### 2. INTRODUCTION

BNT162b2 is an RNA-based COVID-19 vaccine that is currently in use via either emergency (temporary) use or conditional marketing authorizations in approximately 70 countries for the prevention of COVID-19 in individuals ≥16 years of age. BNT162b2 received first temporary authorization for emergency supply under regulation 174 in the UK on 01 December 2020 and is currently authorized for emergency use in 30 countries. BNT162b2 received first regulatory conditional marketing authorization approval in Switzerland on 19 December 2020 and is currently conditionally approved in 40 countries.

#### 2.1. Study Rationale

The purpose of this study is to demonstrate that the immune response induced by the refrigerator-stable lyophilized formulation of BNT162b2 is noninferior to the frozen-liquid formulation of BNT162b2 in MDVs, and to describe the safety and tolerability of these different vaccine formulations in healthy adults, thereby supporting refrigerated storage and distribution at commercial scale. The study will also describe the safety and immunogenicity of frozen-liquid BNT162b2 with LNP size at the upper end of specification and RTU BNT162b2.

Current clinical and EUA specifications for LNP size for the frozen-liquid formulation are 40 to 180 nm and 40 to 120 nm, respectively. Clinical experience, however, is limited to LNP size in the range 59 to 74 nm, based on lots used in the clinical studies already conducted. Hence, an exploratory study arm is being included to better understand the impact of LNP size, using a lot with LNP size close to the upper specification boundary (without any significant impact on other quality attributes). The immediate manufacturing precursor of the lyophilized formulation is the RTU. An exploratory study arm is included to describe the safety and immunogenicity of the RTU (ie, precursor prior to the lyophilization step).

The primary immunogenicity analysis demonstrated that the immune response elicited by the lyophilized formulation did not meet the noninferiority criteria compared to the frozen-liquid formulation of BNT162b2. As a result, for the benefit of the participants, all study participants who received 2 doses of the lyophilized formulation will be offered an additional vaccine dose, using the 30-µg dose of the frozen-liquid formulation of BNT162b2.

#### 2.2. Background

In December 2019, a pneumonia outbreak of unknown cause occurred in Wuhan, China. In January 2020, it became clear that a novel coronavirus (2019-nCoV) was the underlying cause. Later in January, the genetic sequence of the 2019-nCoV became available to the WHO and the public (MN908947.3), and the virus was categorized in the *Betacoronavirus* subfamily. By sequence analysis, the phylogenetic tree revealed a closer relationship to SARS virus isolates than to another coronavirus infecting humans, the MERS virus.<sup>1,2</sup>

The outbreak was declared a Public Health Emergency of International Concern on 30 January 2020.<sup>3</sup> On 12 February 2020, the virus was officially named as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), and the WHO officially named the disease caused by SARS-CoV-2 as coronavirus disease 2019 (COVID-19).<sup>3</sup> SARS-CoV-2

infections and the resulting disease, COVID-19, have spread globally and on 11 March 2020, the WHO characterized the COVID-19 outbreak as a pandemic.<sup>4</sup> On 08 January 2021, The Center for Systems Science and Engineering at Johns Hopkins University reported more than 88 million cases globally, with over 1.9 million deaths from 191 countries. The United States has reported more than 21.6 million cases and over 366,000 deaths.<sup>5</sup>

Since fall of 2020, the incidence of COVID-19 illnesses is increasing dramatically in many northern hemisphere countries, including the United States, France, Germany, Italy, and the United Kingdom, raising the specter that as temperatures have fallen and the "respiratory virus season" has started, cases may dramatically increase, potentially overwhelming healthcare infrastructures. This possibility highlights the importance of developing a COVID-19 vaccine as quickly as possible while ensuring that all safety measures are met.

A prophylactic, RNA-based SARS-CoV-2 vaccine provides one of the most flexible and fastest approaches available to immunize against the emerging virus.<sup>6,7</sup> In an attempt to prevent the spread of disease and to control the pandemic, numerous COVID-19 vaccine candidates are in development.

The development of an RNA-based vaccine encoding a viral antigen, which is then expressed by the vaccine recipient as a protein capable of eliciting protective immune responses, provides significant advantages over more traditional vaccine approaches. Unlike live attenuated vaccines, RNA vaccines do not carry the risks associated with infection and may be given to people who cannot be administered live virus (eg, pregnant women and immunocompromised persons). RNA-based vaccines are manufactured via a cell-free in vitro transcription process, which allows an easy and rapid production and the prospect of producing high numbers of vaccination doses within a shorter time period than achieved with traditional vaccine approaches. This capability is pivotal to enable the most effective response in outbreak scenarios.<sup>6,7</sup>

BNT162b2 is a SARS-CoV-2–RNA-LNP vaccine based on a platform of modRNA with blunted innate immune sensor–activating capacity and augmented expression encoding P2 S.

#### 2.2.1. Clinical Overview

Study C4591001 (NCT04368728) is an ongoing Phase 1/2/3 trial in ~44,000 participants designed to generate safety, tolerability, immunogenicity, and efficacy data from a novel RNA-based vaccine candidate.<sup>8</sup> The trial is being conducted in a heterogeneous study population: eligible participants ≥12 years of age, healthy participants, including those participants with stable chronic medical conditions, including HIV-, HCV-, and HBV-positive participants. The study consists of 2 parts: Phase 1: to identify the preferred vaccine candidate (BNT162b1 or BNT162b2) and dose level (10 μg, 20 μg, 30 μg, or 100 μg [for BNT162b1]); Phase 2/3: an expanded-cohort and efficacy part for the selected vaccine candidate (BNT162b2). BNT162b2 was selected from the Phase 1 part of this study based on the overall safety, tolerability, and immunogenicity. In a mid-November 2020 analysis of 36,621 participants randomized 1:1 to vaccine or placebo who were included in the per-protocol efficacy analysis population of participants without evidence of SARS-CoV-2 infection prior to 7 days after completion of the vaccination schedule, efficacy in preventing

confirmed COVID-19 occurring at least 7 days after the second dose of vaccine was 95.0%, with 8 COVID-19 cases in the active vaccine group and 162 COVID-19 cases in the placebo group. Subgroup analyses of the primary efficacy endpoint showed similar efficacy point estimates across age groups, sexes, racial and ethnic groups, and participants with medical comorbidities associated with high risk of severe COVID-19. Secondary efficacy analyses suggested benefit of the vaccine in preventing severe COVID-19, in preventing COVID-19 following the first dose, and in preventing COVID-19 in individuals with prior SARS-CoV-2 infection, although available data for these outcomes did not allow for firm conclusions.

Safety data from approximately 38,000 participants at least 16 years of age randomized 1:1 to vaccine or placebo with a median of 2 months of follow-up after the second dose suggest a favorable safety profile. Available safety data from all participants enrolled through the 14 November 2020 data cutoff (N=43,252, which includes late enrollment of additional adolescent and adult participants) were consistent with the safety profile for the approximately 38,000 participants with a median follow-up of 2 months and also did not raise specific safety concerns.<sup>9</sup>

The most common solicited adverse reactions were injection site reactions (84.1%), fatigue (62.9%), headache (55.1%), muscle pain (38.3%), chills (31.9%), joint pain (23.6%), and fever (14.2%); severe adverse reactions occurred in 0.0% to 4.6% of participants, were more frequent after Dose 2 than after Dose 1, and were generally less frequent in participants  $\geq$ 55 years of age ( $\leq$ 2.8%) as compared to younger participants ( $\leq$ 4.6%). The frequency of SAEs was low (<0.5%), without meaningful imbalances between study arms. Among nonserious unsolicited AEs, there was a numerical imbalance of 4 cases of Bell's palsy in the active vaccine group compared with no cases in the placebo group, though the 4 cases in the active vaccine group do not represent a frequency above that expected in the general population. Otherwise, there were no notable patterns or numerical imbalances between vaccine groups for specific categories of nonserious AEs (including other neurologic, neuroinflammatory, and thrombotic events) that would suggest a causal relationship to BNT162b2. With the exception of more frequent, generally mild to moderate reactogenicity in participants <55 years of age, the safety profile of BNT162b2 was generally similar across age groups, sexes, ethnic and racial groups, participants with or without medical comorbidities, and participants with or without evidence of prior SARS-CoV-2 infection at enrollment.9

In the C4591001 study, the Phase 1 population included healthy participants 18 through 55 and 65 through 85 years of age. Enrollment in Phase 1 is complete and, although follow-up continues, the available safety data from Phase 1 participants show that BNT162b2 reactogenicity, AEs, and laboratory results were consistent with those commonly associated with vaccination. The observed reactogenicity was generally mild or moderate (primarily pain at the injection site) and short-lived. The local reactions tended to be more frequent after the second dose. There was no redness or swelling reported by participants in the 65- through 85-year age group who received BNT162b2.<sup>10</sup>

Regarding systemic events, 17% of the 18- through 55-year age group and 8% of those in the 65- through 85-year age group reported fever (≥38.0°C to 38.9°C) after the second dose of

30 µg of BNT162b2. Severe systemic events (fatigue, headache, chills, muscle pain, and joint pain) were reported in small numbers of younger recipients of this vaccine candidate, but no severe systemic events were reported in older recipients, and there were no Grade 4 systemic events reported.<sup>10</sup>

No unexpected AEs or SAEs were reported. Through 1 month after receipt of the second vaccination, AEs that were considered by investigators to be related to the study intervention were reported in 25% of participants 18 through 55 years of age who received 30 µg of BNT162b2; no AEs were reported by the older population who received the same dose. <sup>10</sup>

The available immunogenicity data from Phase 1 participants show that BNT162b2 induced a robust IgG-binding response to S1 and a SARS-CoV-2–neutralizing response. Immunogenicity substantially increased following the second dose of vaccine. BNT162b2 induces a strong antigen-specific Th 1–skewed CD4+ response and a strong antigen-specific CD8+ response.

Based on the safety, tolerability, and immunogenicity data generated from Phase 1, the vaccine candidate selected for the Phase 2/3 part of the study was BNT162b2 at a dose of 30  $\mu$ g. This phase of the study is currently ongoing and is evaluating the efficacy of the study intervention.

The Phase 2/3 portion of C4591001 was initiated in 18- through 85-year-old adults but was amended in September 2020 to include participants ≥16 years of age. It is intended that a minimum of 40% of participants will be in the >55-year stratum. A further protocol amendment in October 2020 added a stratum of 2000 participants (1000 active vaccine) 12 through 15 years of age. The first 360 participants in the Phase 2/3 part of the study will be considered the Phase 2 segment but will also contribute to the efficacy endpoint.

There are 2 primary efficacy endpoints in the Phase 2/3 part of the study. The first is to evaluate the efficacy of prophylactic BNT162b2 against confirmed COVID-19 in participants without evidence of infection before vaccination and the second is to evaluate the efficacy of prophylactic BNT162b2 against confirmed COVID-19 in participants regardless of evidence of infection before vaccination. Cases of COVID-19 are defined by the presence of specified symptoms plus an NAAT for SARS-CoV-2 at least 7 days following the second dose of vaccine. Effectiveness in 12- to 15-year-old participants will be inferred by immune noninferiority to that in 16- to 25-year-old participants based on SARS-CoV-2—neutralizing GMTs.

The primary safety objective includes definition of the safety profile of prophylactic BNT162b2 in the first 360 participants in the Phase 2 population, in all participants randomized in Phase 2/3, and in 12- to 15-year-old participants. Reactogenicity will be assessed by e-diary in all participants in Phase 1, in at least 6000 participants in Phase 2/3, and in all participants 12 through 15 years of age.

The scale of the BNT162b2 manufacturing has been increased to support future supply. Therefore, in the C4591001 Phase 2/3 phase of the study, BNT162b2 generated using the

manufacturing process supporting an increased supply ("Process 2") was administered to approximately 250 participants 16 through 55 years of age, per lot.

The currently available safety and immunogenicity data are presented in the BNT162 IB. 11

#### 2.3. Benefit/Risk Assessment

There is an ongoing global pandemic of COVID-19 and, based on the data available from the C4591001 study, multiple temporary or emergency use authorizations and conditional marketing authorizations have been granted for BNT162b2. The available safety and immunogenicity data from the ongoing Pfizer/BioNTech clinical trial combined with available nonclinical data with BNT162 vaccines, and data from nonclinical studies and clinical trials with the same or related RNA components, or antigens, support a favorable benefit/risk profile and support continued clinical development of BNT162b2.

In the C4591001 study, BNT162b2 has been shown to elicit increased local and systemic adverse reactions as compared to those in the placebo arm, usually lasting a few days. The most common solicited adverse reactions were injection site reactions (84.1%), fatigue (62.9%), headache (55.1%), muscle pain (38.3%), chills (31.9%), joint pain (23.6%), and fever (14.2%). Adverse reactions characterized as reactogenicity were generally mild to moderate. The number of participants reporting hypersensitivity-related AEs was numerically higher in the active vaccine group compared with the placebo group (137 [0.63%] vs 111 [0.51%]). Severe adverse reactions occurred in 0.0% to 4.6% of participants, were more frequent after Dose 2 than after Dose 1, and were generally less frequent in older adults (>55 years of age) (<2.8%) as compared to younger participants (≤4.6%). Among reported unsolicited AEs, lymphadenopathy occurred much more frequently in the active vaccine group than the placebo group and is plausibly related to vaccination. SAEs, while uncommon (<1.0%), represented medical events that occur in the general population at similar frequency as observed in the study.

No specific safety concerns were identified in subgroup analyses by age, race, ethnicity, medical comorbidities, or prior SARS-CoV-2 infection. Although participants 16 through 17 years of age were enrolled in the Phase 3 trial, safety data for this age group are limited. However, available data are consistent with the safety profile in the adult population, and it is biologically reasonable to extrapolate the greater safety experience in adults, in particular younger adults, to the oldest pediatric age group of 16 through 17 years. The potential risks are based on the observed safety profile to date, which shows mostly mild reactogenicity, low incidence of severe or serious events, and no clinically concerning safety observations. The preponderance of severe cases of COVID-19 in the placebo group relative to the BNT162b2 group (9 of 10) suggests no evidence of VAED. Continued clinical investigation is justified given:

the urgent need to optimize storage and distribution of a COVID-19 vaccine on a
wide scale using a lyophilized formulation that will be stable at standard refrigerator
temperatures,

- the threat posed by the increasing number of globally distributed outbreaks of SARS-CoV-2 infection,
- the potential of the BioNTech platform of RNA-based vaccines to rapidly deliver high numbers of vaccine doses in a single production campaign.

More detailed information about the known and expected benefits and risks and reasonably expected AEs of BNT162b2 may be found in the IB, which is the SRSD for this study.

# 2.3.1. Risk Assessment

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Study | Study Intervention: BNT162b2 RNA-Based COVID-19 Vaccine | |
| Local and systemic reactions to the vaccine may occur (injection site redness, injection site swelling, and injection site pain, fever, fatigue, headache, chills, muscle pain, and joint pain) following vaccination. | These are common adverse reactions seen with other vaccines as well as the COVID-19 vaccine. The most common events reported in Study C4591001 were mild to moderate pain at the injection site, fatigue, and headache. | <ul> <li>The study employs the use of a reactogenicity e-diary to monitor local reactions and systemic events in real time.</li> <li>All study participants will be observed for at least 30 minutes after vaccination.</li> </ul> |
| Safety profile of a novel vaccine not yet fully characterized. Adverse reactions (risks) identified from the postauthorization safety data include: Anaphylaxis, other hypersensitivity reactions (eg, rash, pruritus, urticaria, angioedema), pain in extremity (injected arm). | Data available from Study C4591001 showed low incidence of severe or serious events, and no clinically concerning safety observations across the safety population and within demographic subgroups based on age, sex, race/ethnicity, country, and baseline SARS-CoV-2 status. Postauthorization safety data surveillance has confirmed the safety profile observed in C4591001 and has resulted in identification of some additional adverse reactions (risks) as noted in this table. | <ul> <li>Collection of AE and SAE reports from signing of the ICD through 1 month after the second dose of vaccine.</li> <li>DMC throughout the study to review all safety data.</li> <li>All participants will be observed for at least 30 minutes after vaccination.</li> </ul> |
| Potential for COVID-19 enhancement. | Disease enhancement has been seen following vaccination with RSV, feline coronavirus, and Dengue virus vaccines. No evidence of disease enhancement has been seen in large-scale clinical study of BNT162b2 in humans or in postauthorization surveillance. | <ul> <li>Eligibility criteria will exclude any participants who have had a previous clinical (signs/symptoms only) or microbiological (signs/symptoms and positive SARS-CoV-2 NAAT result) diagnosis of COVID-19. This will minimize the low risk of potential disease enhancement and ensure that the immune response evaluated in the study is not impacted by serological changes due to previous COVID-19 disease.</li> <li>Monitoring for cases of COVID-19 developing during the study, which will be reported as AESIs.</li> </ul> |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Study Procedures | | |
| Participants will be required to attend healthcare facilities during the global SARS-CoV-2 pandemic. | Without appropriate social distancing and PPE, there is a potential for increased exposure to SARS-CoV-2. | <ul> <li>Pfizer will work with sites to ensure an appropriate COVID-19 prevention strategy.</li> <li>The study will include monitoring for cases of COVID-19 developing during the study, which will be reported as AESIs.</li> </ul> |
| Venipuncture will be performed during the study. | There is the risk of bleeding, bruising, hematoma formation, and infection at the venipuncture site. | Only appropriately qualified personnel will obtain the blood draw. |
| Very rare cases of anaphylaxis, myocarditis, and pericarditis have been reported after EUA in recipients of BNT162b2 | Anaphylaxis: The estimated rate is 5.0 per million doses administered. Myocarditis and pericarditis: Very rare cases of myocarditis and pericarditis have been reported following vaccination with mRNA COVID-19 vaccines. Typically, these cases have occurred more often in younger men and after the second dose of the vaccine and within 14 days after vaccination. These are generally mild cases and individuals tend to recover within a short time following standard treatment and rest. Healthcare professionals should be alert to the signs and symptoms of myocarditis and pericarditis in vaccine recipients. | Specific reference to these risks is made within the ICD, with instruction to contact a healthcare professional if a case is suspected. For anaphylaxis, there is an on-site observation period of 30-minute after vaccination. Instructions for handling suspected cases of myocarditis and pericarditis are found in Section 8.13. |

#### 2.3.2. Benefit Assessment

Benefits to individual participants may include:

- Receipt of an efficacious or potentially efficacious COVID-19 vaccine during a global pandemic
- Access to COVID-19 diagnostic testing
- Contributing to research to help others in a time of global pandemic

# 2.3.3. Overall Benefit/Risk Conclusion

Taking into account the measures taken to minimize risks to participants participating in this study, the potential risks identified in association with BNT162b2 are justified by the anticipated benefits that may be afforded to healthy participants.

# 3. OBJECTIVES, ESTIMANDS, AND ENDPOINTS

| Objectives | Estimands | Endpoints |
|---|---|---|
| Primary Immunogenicity | | |
| To demonstrate that the immune response induced by lyophilized BNT162b2 in SDVs is noninferior to the immune response induced by frozenliquid BNT162b2 in MDVs in participants without evidence of SARS-CoV-2 infection during the study | In participants complying with the key protocol criteria (evaluable participants): • GMR of lyophilized formulation in SDVs relative to frozen-liquid formulation in MDVs 1 month after Dose 2 | Full-length S-binding IgG levels |
| | Primary Safety | |
| To evaluate the safety of<br>BNT162b2 when administered<br>on a 2-dose schedule in healthy<br>adults 18 through 55 years of<br>age | In participants receiving at least 1 dose of study intervention from each vaccine group, the percentage of participants reporting: • Local reactions for up to 7 days following each dose • Systemic events for up to 7 days following each dose • AEs and SAEs from Dose 1 through 1 month after Dose 2 | <ul> <li>Local reactions (pain at the injection site, redness, and swelling)</li> <li>Systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain)</li> <li>AEs</li> <li>SAEs</li> </ul> |
| Secondary Immunogenicity | | |
| To describe the immune responses induced by lyophilized BNT162b2 in SDVs and frozen-liquid BNT162b2 in MDVs | In evaluable participants from each vaccine group: • GMCs at baseline (before Dose 1) and 1 month after Dose 2 • GMFR from baseline (before Dose 1) to 1 month after Dose 2 | Full-length S-binding IgG levels |


| Objectives | Estimands | Endpoints |
|---|---|---|
| | Exploratory | |
| To describe the immune responses induced by frozen-liquid BNT162b2 with LNP size at the upper end of specification and RTU BNT162b2 in participants without evidence of SARS-CoV-2 infection during the study | In evaluable participants: • GMR of frozen-liquid BNT162b2 with LNP size at the upper end of specification relative to frozen-liquid BNT162b2 in MDVs 1 month after Dose 2 | Full-length S-binding IgG<br>levels and/or SARS-CoV-2<br>neutralizing titers |
| To describe the immune responses induced by frozen-liquid BNT162b2 with LNP size at the upper end of specification and RTU BNT162b2 | In evaluable participants from each vaccine group: • GMCs and/or GMTs at baseline (before Dose 1) and 1 month after Dose 2 • GMFR from baseline (before Dose 1) to 1 month after Dose 2 | Full-length S-binding IgG<br>levels and/or SARS-CoV-2<br>neutralizing titers |
| To describe the safety profile of frozen-liquid BNT162b2 formulation when given as a third dose to participants who originally received 2 doses of the lyophilized formulation of BNT162b2 | In participants who originally received 2 dose series of the lyophilized formulation of BNT162b2: • Local reactions for up to 7 days following third dose • Systemic events for up to 7 days following third dose • AEs from Dose 3 to 1 month after Dose 3 • SAEs from Dose 3 to 1 month after Dose 3 | <ul> <li>Local reactions (pain at the injection site, redness, and swelling)</li> <li>Systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain)</li> <li>AEs</li> <li>SAEs</li> </ul> |
| To describe the immune response elicited by frozen-liquid BNT162b2 formulation when given as third dose following a primary series of lyophilized BNT162b2 | In evaluable participants who originally received 2 dose series of the lyophilized formulation of BNT162b2 GMFR from prior to Dose 3 to 1 month after Dose 3 GMCs and/or GMTs at baseline, at 1 month after Dose 2, prior to Dose 3 and 1 month after Dose 3 | Full-length S-binding IgG<br>levels and/or SARS-CoV-2<br>neutralizing titers |

#### 4. STUDY DESIGN

# 4.1. Overall Design

This is a Phase 3, randomized, observer-blind study to evaluate the safety, tolerability, and immunogenicity of multiple formulations of BNT162b2, an RNA-based COVID-19 vaccine, administered on a 2-dose schedule in healthy adults 18 through 55 years of age. The study will be conducted in the US with potential to expand to other countries.

In Part 1, participants will receive either lyophilized BNT162b2 in SDVs or frozen-liquid BNT162b2 in MDVs. In Part 2, participants will receive either frozen-liquid BNT162b2 with LNP size at the upper end of specification or RTU BNT162b2. In Part 1, participants will be randomized in a 1:1 ratio to 1 of the 2 groups (lyophilized SDV or frozen-liquid MDV control for lyophilized SDV). Separately, in Part 2, participants will be randomized in a 1:1 ratio to 1 of the 2 groups (frozen-liquid BNT162b2 with LNP size at the upper end of specification or RTU BNT162b2). The duration of the study for each participant will be approximately 2 months. Approximately 550 participants will be randomly assigned to either lyophilized SDV or frozen-liquid MDV control for lyophilized SDV; separately, approximately 60 participants will be randomly assigned to receive either frozen-liquid BNT162b2 with LNP size at the upper end of specification or RTU BNT162b2, for a total of approximately 610 randomized participants. It is expected that approximately 488 evaluable participants will complete the study, based on a 20% nonevaluable rate.

Updates as part of protocol amendment 2:

All participants who originally received 2 doses of the lyophilized formulation of BNT162b2 will be offered the opportunity to receive a third dose with the current frozen-liquid formulation of BNT162b2. Those participants who accept the offer of receiving third dose will have 2 additional visits as described in Section 1.3.1. The study duration will be extended for 1 additional month for those participants who accept the offer of receiving a third dose.

#### 4.2. Scientific Rationale for Study Design

This study contains assessments that could be considered standard for a vaccine noninferiority study. Blood samples taken for immunogenicity will establish the level of immune response elicited by each formulation to provide the necessary data to meet the primary endpoint of the study. Immunogenicity will be assessed by the full-length S-binding IgG assay. To establish if a participant has asymptomatic SARS-CoV-2 infection, nasal swabs for SARS-CoV-2 nucleic acid amplification testing (ie, NAAT) and blood samples to measure N-binding antibody levels will be taken. A positive result on either test will result in the immunogenicity data from that participant being excluded from the evaluable portion of the study population. All reactogenicity and safety assessments are standard for a study of this nature.

This study will not include a placebo, as the aim and design of this study are not to demonstrate efficacy.

Human reproductive safety data are not available for BNT162b2, but there is no suspicion of human teratogenicity based on the intended mechanism of action of the compound. Therefore, the use of a highly effective method of contraception is required (see Appendix 4).

#### 4.3. Justification for Dose

Based on data from the Phase 1 component of clinical trial C4591001 and available nonclinical data, the modRNA BNT162b2 vaccine candidate was selected at a dose of 30  $\mu$ g for Phase 2/3 evaluation of safety, immunogenicity, and efficacy. This is the dose that has shown to be effective and has been authorized for temporary or emergency use.

Update based on protocol amendment 2:

The primary immunogenicity analysis demonstrated that the immune response elicited by the lyophilized formulation did not meet the noninferiority criteria compared to the frozen-liquid formulation. Therefore, all study participants who received 2 doses of the lyophilized formulation will be offered an additional 30-ug dose of the frozen-liquid formulation.

#### 4.4. End of Study Definition

A participant is considered to have completed the study if he/she has completed all phases of the study, including the last visit.

The end of the study is defined as the date of the last visit of the last participant in the study.

#### 5. STUDY POPULATION

This study can fulfill its objectives only if appropriate participants are enrolled. The following eligibility criteria are designed to select participants for whom participation in the study is considered appropriate. All relevant medical and nonmedical conditions should be taken into consideration when deciding whether a particular participant is suitable for this protocol.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

#### 5.1. Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

#### Age and Sex:

- 1. Male or female participants between the ages of 18 and 55 years, inclusive, at Visit 1 (Day 1).
  - Refer to Section 10.4 for reproductive criteria for male (Section 10.4.1) and female (Section 10.4.2) participants.

#### **Type of Participant and Disease Characteristics:**

2. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

3. Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

Note: Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included.

#### **Informed Consent:**

- 4. Capable of giving personal signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.
- 5. For Dose 3: Participants who received BOTH doses of the lyophilized formulation of BNT162b2 as part of the initial study.

#### 5.2. Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

#### **Medical Conditions:**

- 1. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
- 2. Known infection with HIV, HCV, or HBV.
- 3. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
- 4. Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID-19.
- 5. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
- 6. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
- 7. Women who are pregnant or breastfeeding.

# **Prior/Concomitant Therapy:**

8. Previous vaccination with any coronavirus vaccine.

- 9. Receipt of medications intended to prevent COVID-19.
- 10. Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (if systemic corticosteroids are administered for ≥14 days at a dose of ≥20 mg/day of prednisone or equivalent), eg, for cancer or an autoimmune disease, or planned receipt throughout the study. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
- 11. Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.

#### **Prior/Concurrent Clinical Study Experience:**

- 12. Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
- 13. Previous participation in other studies involving study intervention containing LNPs.

#### **Other Exclusions:**

14. Investigator site staff or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

#### 5.3. Lifestyle Considerations

#### **5.3.1.** Contraception

The investigator or his or her designee, in consultation with the participant, will confirm that the participant has selected an appropriate method of contraception for the individual participant and his or her partner(s) from the permitted list of contraception methods (see Section 10.4.4) and will confirm that the participant has been instructed in its consistent and correct use.

At time points indicated in the SoA, the investigator or designee will inform the participant of the need to use highly effective contraception consistently and correctly and document the conversation and the participant's affirmation in the participant's chart (participants need to affirm their consistent and correct use of at least 1 of the selected methods of contraception). In addition, the investigator or designee will instruct the participant to call immediately if the selected contraception method is discontinued or if pregnancy is known or suspected in the participant or partner.

#### 5.4. Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently randomly assigned to study intervention. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the CONSORT publishing requirements and to respond to queries from regulatory

authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any SAEs.

Individuals who do not meet the criteria for participation in this study (screen failure) may be rescreened under a different participant number.

# 5.5. Criteria for Temporarily Delaying Enrollment/Randomization/Study Intervention Administration

The following conditions are temporary or self-limiting and a participant may be vaccinated once the condition(s) has/have resolved and no other exclusion criteria are met. Participants meeting these criteria at Vaccination 1 will be considered screen failures if enrollment has closed once the condition(s) has/have resolved.

- 1. Current febrile illness (body temperature ≥100.4°F [≥38.0°C]) or other acute illness within 48 hours before study intervention administration. This includes current symptoms that could represent a potential COVID-19 illness:
  - New or increased cough;
  - New or increased shortness of breath;
  - Chills;
  - New or increased muscle pain;
  - New loss of taste/smell;
  - Sore throat:
  - Diarrhea;
  - Vomiting.
- 2. Receipt of any seasonal or pandemic influenza vaccine within 14 days, or any other nonstudy vaccine within 28 days, before study intervention administration.
- 3. Anticipated receipt of any seasonal or pandemic influenza vaccine within 14 days, or any other nonstudy vaccine within 28 days, after study intervention administration.
- 4. Receipt of short-term (<14 days) systemic corticosteroids. Study intervention administration should be delayed until systemic corticosteroid use has been discontinued for at least 28 days. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.

#### 6. STUDY INTERVENTION

Study intervention is defined as any investigational intervention(s), marketed product(s), placebo, medical device(s), or study procedure(s) intended to be administered to a study participant according to the study protocol.

For the purposes of this protocol, study intervention refers to BNT162b2, an RNA-based vaccine for immunization against COVID-19. One of 3 versions of BNT162b2 (lyophilized, frozen-liquid, or RTU) will be administered to each participant. The study will evaluate a 2-dose (separated by 21 days) schedule in healthy adults 18 through 55 years of age.

# 6.1. Study Intervention(s) Administered

| Intervention Name | BNT162b2<br>(BNT162 RNA-LNP vaccine utilizing modRNA) | BNT162b2<br>(BNT162 RNA-LNP vaccine utilizing modRNA) | BNT162b2<br>(BNT162 RNA-LNP<br>vaccine utilizing<br>modRNA) |
|---|---|---|---|
| Arm Name<br>(group of participants<br>receiving a specific<br>vaccine or no vaccine) | Frozen-liquid MDV | Lyophilized SDV | RTU SDV |
| Type | Vaccine | Vaccine | Vaccine |
| <b>Dose Formulation</b> | modRNA | modRNA | modRNA |
| Dosage Level | 30 μg | 30 μg | 30 μg |
| Route of Administration | Intramuscular injection | Intramuscular injection | Intramuscular injection |
| Use | Experimental | Experimental | Experimental |
| IMP or NIMP | IMP | IMP | IMP |
| Sourcing | Provided centrally by the sponsor | Provided centrally by the sponsor | Provided centrally by the sponsor |
| Packaging and<br>Labeling | Study intervention will be provided in a glass vial. Each vial will be labeled as required per country requirement. | Study intervention will be provided in a glass vial. Each vial will be labeled as required per country requirement. | Study intervention will be provided in a glass vial. Each vial will be labeled as required per country requirement. |

#### 6.1.1. Administration

Participants will receive 1 dose of study intervention as randomized at each vaccination visit (Visits 1 and 2) separated by 21 days in accordance with the study's SOA. Full details are described in the IP manual.

Participants who originally received 2 doses of the lyophilized formulation of BNT162b2 will be offered the opportunity to receive an additional dose of the frozen-liquid formulation of BNT162b2 at least 90 days after Dose 2.

Study intervention should be administered intramuscularly into the deltoid muscle, preferably of the nondominant arm, by an **unblinded** administrator.

Standard vaccination practices must be observed and vaccine must not be injected into blood vessels. Appropriate medication and other supportive measures for management of an acute hypersensitivity reaction should be available in accordance with local guidelines for standard immunization practices.

Administration of study interventions should be performed by an appropriately qualified, GCP-trained, and vaccine-experienced member of the study staff (eg, physician, nurse, physician's assistant, nurse practitioner, pharmacist, or medical assistant) as allowed by local, state, and institutional guidance.

Study intervention administration details will be recorded on the CRF.

### 6.2. Preparation/Handling/Storage/Accountability

- 1. The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study interventions received and any discrepancies are reported and resolved before use of the study intervention.
- 2. Only participants enrolled in the study may receive study intervention and only authorized site staff may supply or administer study intervention. All study interventions must be stored in a secure, environmentally controlled, and monitored (manual or automated recording) area in accordance with the labeled storage conditions with access limited to the investigator and authorized site staff. The temperature of all locations where study intervention is stored at a clinical site must be monitored continuously. At a minimum, daily minimum and maximum temperatures for all site storage locations must be documented and available upon request. Data for nonworking days must indicate the minimum and maximum temperatures since previously documented for all site storage locations upon return to business.
- 3. Any excursions from the study intervention label storage conditions should be reported to Pfizer upon discovery along with any actions taken. The site should actively pursue options for returning the study intervention to the storage conditions described in the labeling, as soon as possible. Once an excursion is identified, the study intervention must be quarantined and not used until Pfizer provides permission to use the study intervention. Specific details regarding the definition of an excursion and information the site should report for each excursion will be provided to the site in the IP manual.
- 4. Any storage conditions stated in the SRSD will be superseded by the storage conditions stated on the label.
- 5. Study interventions should be stored in their original containers.
- 6. See the IP manual for storage conditions of the study intervention.

- 7. The investigator, institution, or the head of the medical institution (where applicable) is responsible for study intervention accountability, reconciliation, and record maintenance (ie, receipt, reconciliation, and final disposition records), such as the IPAL or sponsor-approved equivalent. All study interventions will be accounted for using a study intervention accountability form/record.
- 8. Further guidance and information for the final disposition of unused study interventions are provided in the IP manual. All destruction must be adequately documented. If destruction is authorized to take place at the investigator site, the investigator must ensure that the materials are destroyed in compliance with applicable environmental regulations, institutional policy, and any special instructions provided by Pfizer.

Upon identification of a product complaint, notify the sponsor within 1 business day of discovery as described in the IP manual.

#### 6.2.1. Preparation and Dispensing

See the IP manual for instructions on how to prepare the study intervention for administration. Study intervention should be prepared and dispensed by an appropriately qualified and experienced member of the study staff (eg, physician, nurse, physician's assistant, nurse practitioner, pharmacy assistant/technician, or pharmacist) as allowed by local, state, and institutional guidance. A second staff member will verify the preparation and dispensing.

Study intervention will be prepared by qualified unblinded site personnel according to the IP manual. The study intervention will be administered in such a way as to ensure the participants remain blinded.

Requirements for site personnel to be blinded for the Dose 3 preparation are not applicable.

#### 6.3. Measures to Minimize Bias: Randomization and Blinding

#### 6.3.1. Allocation to Study Intervention

Allocation (randomization) of participants to vaccine groups will proceed through the use of an IRT system (IWR). The site personnel (study coordinator or specified designee) will be required to enter or select information including but not limited to the user's ID and password, the protocol number, and the participant number. The site personnel will then be provided with a vaccine assignment and randomization number. The IRT system will provide a confirmation report containing the participant number, randomization number, and study intervention allocation assigned. The confirmation report must be stored in the site's files.

The study-specific IRT reference manual and IP manual will provide the contact information and further details on the use of the IRT system.

#### **6.3.2.** Blinding of Site Personnel

In this observer-blinded study, the study staff receiving, storing, dispensing, preparing, and administering the study interventions will be unblinded. All other study and site personnel, including the investigator, investigator staff, and participants, will be blinded to study intervention assignments. In particular, the individuals who evaluate participant safety will be blinded.

The PI will assign the responsibility of the unblinded dispensers/administrators to persons who will not participate in the evaluation of any study participant. To ensure adequate coverage, at least 2 unblinded dispensers/administrators will be assigned per site. Members of the study site staff or clinic pharmacy should fulfill these roles. Contact between the unblinded dispensers and study participants should be kept to a minimum. The investigator, study coordinator, and any site staff other than the unblinded dispensers/administrators must not be allowed to know the study intervention assigned to any study participant and must not be allowed to see the study intervention container contents. Once the study intervention has been prepared, there is no difference in the physical appearance of the BNT162b2 formulations. In the event of a Quality Assurance audit, the auditor(s) will be allowed access to unblinded study intervention records at the site(s) to verify that randomization/dispensing has been done accurately.

Update based on protocol amendment 2:

After the complete data through 1 month after Dose 2 for Part 1 participants were available, the database for Part 1 was released and unblinded for the study team to perform the statistical analyses specified for Part 1. Additionally, site staff and study participants were also unblinded to participants' vaccine allocation.

#### 6.3.3. Blinding of the Sponsor

The majority of sponsor staff will be blinded to study intervention allocation. All laboratory testing personnel performing serology assays will remain blinded to study intervention assigned/received throughout the study. The following sponsor staff, who will have no part in the blinded conduct of the study, will be unblinded (further details will be provided in a data blinding plan):

- Those study team members who are involved in ensuring that protocol requirements for study intervention preparation, handling, allocation, and administration are fulfilled at the site will be unblinded for the duration of the study (eg, unblinded study manager, unblinded clinical research associate).
- Unblinded clinician(s) who are not direct members of the study team and will not
  participate in any other study-related activities will review unblinded protocol
  deviations.
• After the complete data through 1 month after Dose 2 for Part 1 participants were available, the database for Part 1 was released and unblinded for the study team to perform the statistical analyses specified for Part 1.

## 6.3.4. Breaking the Blind

All study participants will receive BNT162b2; blinding refers only to which vaccine formulation the participant will receive. The IRT will be programmed with blind-breaking instructions. In case of an emergency, the investigator has the sole responsibility for determining if unblinding of a participant's study intervention assignment is warranted. Participant safety must always be the first consideration in making such a determination. If the investigator decides that unblinding is warranted, the investigator should make every effort to contact the sponsor prior to unblinding a participant's vaccine assignment unless this could delay further management of the participant. If a participant's vaccine assignment is unblinded, the sponsor must be notified within 24 hours after breaking the blind. The date and reason that the blind was broken must be recorded in the source documentation and CRF.

The study-specific IRT reference manual and IP manual will provide the contact information and further details on the use of the IRT system.

## 6.4. Study Intervention Compliance

When participants are dosed at the site, they will receive study intervention directly from the investigator or designee, under medical supervision. The date and time of each dose administered in the clinic will be recorded in the source documents and recorded in the CRF. The dose of study intervention and study participant identification will be confirmed at the time of dosing by a member of the study site staff other than the person administering the study intervention.

## 6.5. Concomitant Therapy

The following concomitant medications and vaccinations will be recorded in the CRF:

- All vaccinations received from 28 days prior to study enrollment until the 1-month follow-up visit (Visit 3).
- Additionally, for all participants receiving Dose 3, all vaccinations received from 28 days prior to Visit 101 (Dose 3) until the 1-month follow-up visit (Visit 102).
- Prohibited medications listed in Section 6.5.1 will be recorded, to include start and stop dates, name of the medication, dose, unit, route, and frequency.

#### 6.5.1. Prohibited During the Study

Receipt of the following vaccines and medications during the time periods listed below may exclude a participant from the per-protocol analysis from that point onward and may require vaccinations to be discontinued in that participant; however, it is anticipated that the participant would not be withdrawn from the study (see Section 7). Medications should not be withheld if required for a participant's medical care.


- Unless considered medically necessary, no vaccines other than study intervention should be administered within 28 days before and 28 days after each study vaccination. One exception to this is that seasonal and pandemic influenza vaccine can be given at least 14 days after, or at least 14 days prior to, the administration of study intervention.
- Receipt of chronic systemic treatment with known immunosuppressant medications, or radiotherapy, within 60 days before enrollment through conclusion of the study.
- Receipt of systemic corticosteroids (≥20 mg/day of prednisone or equivalent) for ≥14 days is prohibited from 28 days prior to enrollment through Visit 3 or Visit 102 for those participants receiving Dose 3.
- Receipt of blood/plasma products or immunoglobulins within 60 days before enrollment through conclusion of the study.
- Receipt of any other (nonstudy) coronavirus vaccine at any time prior to or during study participation is prohibited.
- Receipt of prophylactic medications intended to <u>prevent</u> symptoms associated with COVID-19. However, if a participant is taking a medication for another condition, even if it may have such properties, it should not be withheld prior to study vaccination.
- Prophylactic antipyretics and other pain medication to <u>prevent</u> symptoms associated with study intervention administration are not permitted. However, if a participant is taking a medication for another condition, even if it may have antipyretic or pain-relieving properties, it should not be withheld prior to study vaccination.

## 6.5.2. Permitted During the Study

The use of antipyretics and other pain medication to <u>treat</u> symptoms associated with study intervention administration or ongoing conditions is permitted.

Medication other than that described as prohibited in Section 6.5.1 required for treatment of preexisting stable conditions is permitted.

Inhaled, topical, or localized injections of corticosteroids (eg, intra-articular or intrabursal administration) are permitted.

#### 6.6. Dose Modification

Not applicable for this study.

#### 6.7. Intervention After the End of the Study

No intervention will be provided to study participants at the end of the study.

## 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

## 7.1. Discontinuation of Study Intervention

In rare instances, it may be necessary for a participant to permanently discontinue study intervention (definitive discontinuation). Reasons for definitive discontinuation of study intervention include the following: AEs; participant request; investigator request; pregnancy; protocol deviation (including no longer meeting all the inclusion criteria, or meeting 1 or more exclusion criteria\*). In general, unless the investigator considers it unsafe to administer the second dose, or the participant does not wish to receive it, it is preferred that the second dose be administered.

\*A positive SARS-CoV-2 NAAT result without symptoms or a COVID-19 diagnosis (signs/symptoms only or signs/symptoms and a positive SARS-CoV-2 NAAT result) should not result in discontinuation of study intervention. If study intervention (Dose 2) has been delayed per Section 5.5, because of febrile or other acute illness (Item 1 in the list in Section 5.5), and the investigator later diagnoses the signs and symptoms as COVID-19 (with or without a positive SARS-CoV-2 NAAT result), the participant should not be discontinued from any further doses of study intervention.

Note that discontinuation of study intervention does not represent withdrawal from the study. Per the study estimands, if study intervention is definitively discontinued, the participant will remain in the study to be evaluated for safety and immunogenicity. See the SoA for data to be collected at the time of discontinuation of study intervention and follow-up for any further evaluations that need to be completed.

In the event of discontinuation of study intervention, it must be documented on the appropriate CRF/in the medical records whether the participant is discontinuing further receipt of study intervention or also from study procedures, postvaccination study follow-up, and/or future collection of additional information.

## 7.2. Participant Discontinuation/Withdrawal From the Study

A participant may withdraw from the study at any time at his/her own request. Reasons for discontinuation from the study include the following:

- Refused further follow-up;
- Lost to follow-up;
- Death:
- Study terminated by sponsor;
- AEs;
- Participant request;


- Investigator request;
- Protocol deviation.

If a participant does not return for a scheduled visit, every effort should be made to contact the participant. All attempts to contact the participant and information received during contact attempts must be documented in the participant's source document. In any circumstance, every effort should be made to document participant outcome, if possible.

The investigator or his or her designee should capture the reason for withdrawal in the CRF for all participants.

If a participant withdraws from the study, he/she may request destruction of any remaining samples taken and not tested, and the investigator must document any such requests in the site study records and notify the sponsor accordingly.

If the participant withdraws from the study and also withdraws consent (see Section 7.2.1) for disclosure of future information, no further evaluations should be performed and no additional data should be collected. The sponsor may retain and continue to use any data collected before such withdrawal of consent.

Lack of completion of all or any of the withdrawal/early termination procedures will not be viewed as protocol deviations so long as the participant's safety was preserved.

#### 7.2.1. Withdrawal of Consent

Participants who request to discontinue receipt of study intervention will remain in the study and must continue to be followed for protocol-specified follow-up procedures. The only exception to this is when a participant specifically withdraws consent for any further contact with him or her or persons previously authorized by the participant to provide this information. Participants should notify the investigator in writing of the decision to withdraw consent from future follow-up, whenever possible. The withdrawal of consent should be explained in detail in the medical records by the investigator, as to whether the withdrawal is only from further receipt of study intervention or also from study procedures and/or postvaccination study follow-up, and entered on the appropriate CRF page. In the event that vital status (whether the participant is alive or dead) is being measured, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.

#### 7.3. Lost to Follow-up

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to attend a required study visit:

• The site must attempt to contact the participant and reschedule the missed visit as soon as possible and counsel the participant on the importance of maintaining the

assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study;

- Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record;
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.

#### 8. STUDY ASSESSMENTS AND PROCEDURES

The investigator (or an appropriate delegate at the investigator site) must obtain a signed and dated ICD before performing any study-specific procedures.

The full date of birth will be collected to critically evaluate the immune response and safety profile by age.

Study procedures and their timing are summarized in the SoA. Protocol waivers or exemptions are not allowed.

Safety issues should be discussed with the sponsor immediately upon occurrence or awareness to determine whether the participant should continue or discontinue study intervention.

Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.

All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.

Every effort should be made to ensure that protocol-required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances outside the control of the investigator that may make it unfeasible to perform the test. In these cases, the investigator must take all steps necessary to ensure the safety and well-being of the participant. When a protocol-required test cannot be performed, the investigator will document the reason for the missed test and any corrective and preventive actions that he or she has taken to ensure that required processes are adhered to as soon as possible. The study team must be informed of these incidents in a timely manner.

For samples being collected and shipped, detailed collection, processing, storage, and shipment instructions and contact information will be provided to the investigator site prior to initiation of the study.

The total blood sampling volume for individual participants in this study is approximately 40 mL. Additional blood samples may be taken for safety assessments at times specified by Pfizer, provided the total volume taken during the study does not exceed 550 mL during any period of 60 consecutive days.

Per protocol amendment 2, those participants who accept the offer to receive Dose 3 will have an additional approximately 20-mL blood sample collected for immunogenicity assessments at each visit.

## 8.1. Efficacy and/or Immunogenicity Assessments

Serum samples will be obtained for immunogenicity testing at the visits specified in the SoA. The test to be performed will be the SARS-CoV-2 full-length S-binding IgG-level assay. Note that all immunogenicity analyses will be based upon samples analyzed at the central laboratory.

Nasal (midturbinate) swabs at the visits specified in the SoA will be obtained as one of the determinations for participants to be included in the evaluable immunogenicity analysis. These samples will be tested at the central laboratory using an RT-PCR test (Cepheid, an NAAT; FDA approved under EUA) to detect SARS-CoV-2. Another determination for participants to be included in the evaluable immunogenicity analysis is the N-binding antibody assay. Blood samples will be taken at visits specified in the SoA and analyzed at the central laboratory. A positive result on either test will result in the immunogenicity data from that participant being excluded from the evaluable portion of the study population. However, administration of study intervention is not dependent on these test results, which will be available only after the study has ended.

#### 8.1.1. Biological Samples

Blood and nasal swab samples will be used only for scientific research. Each sample will be labeled with a code so that the laboratory personnel testing the samples will not know the participant's identity. Samples that remain after performing assays outlined in the protocol may be stored by Pfizer. Unless a time limitation is required by local regulations or ethical requirements, the samples will be stored for up to 15 years after the end of the study and then destroyed. If allowed by the ICD, stored samples may be used for additional testing to better understand the immune responses to the vaccine(s) under study in this protocol, to inform the development of other products, and/or for vaccine-related assay work supporting vaccine programs. No testing of the participant's genetic material will be performed.

The participant may request that his or her samples, if still identifiable, be destroyed at any time; however, any data already collected from those samples will still be used for this research. The biological samples may be shared with other researchers as long as confidentiality is maintained and no testing of the participant's genetic material is performed.

## 8.2. Safety Assessments

Planned time points for all safety assessments are provided in the SoA. Unscheduled clinical laboratory measurements may be obtained at any time during the study to assess any perceived safety issues.

A clinical assessment, including medical history, will be performed on all participants at their first visit to establish a baseline. Significant medical history and observations from any physical examination, if performed, will be documented in the CRF.

AEs and SAEs are collected, recorded, and reported as defined in Section 8.3.

Acute reactions within the first 30 minutes after administration of the study intervention will be assessed and documented in the AE CRF.

The safety parameters also include reactogenicity e-diary reports of local reactions, systemic events (including fever), and use of antipyretic medication that occur in the 7 days after administration of the study intervention. These prospectively self-collected occurrences of local reactions and systemic events are graded as described in Section 8.2.2.

## 8.2.1. Clinical Safety Laboratory Assessments

Clinical safety laboratory assessments will not be collected in this study.

See Section 10.5, Appendix 5, for suggested actions and follow-up assessments in the event of potential DILI.

## **8.2.2.** Electronic Diary

Participants will be required to complete a reactogenicity e-diary through an application installed on a provisioned device or on the participant's own personal device. All participants will be asked to monitor and record local reactions, systemic events, and antipyretic medication usage for 7 days from the day of administration of the study intervention. The reactogenicity e-diary allows recording of these assessments only within a fixed time window, thus providing the accurate representation of the participant's experience at that time. Data on local reactions and systemic events reported in the reactogenicity e-diary will be transferred electronically to a third-party vendor, where they will be available for review by investigators and the Pfizer clinicians at all times via an internet-based portal.

At intervals agreed to by the vendor and Pfizer, these data will be transferred electronically into Pfizer's database for analysis and reporting. These data do not need to be reported by the investigator in the CRF as AEs.

Investigators (or designee) will be required to review the reactogenicity e-diary data online at frequent intervals as part of the ongoing safety review.

The investigator or designee must obtain stop dates from the participant for any ongoing local reactions, systemic events, or use of antipyretic medication on the last day that the

reactogenicity e-diary was completed. The stop dates should be documented in the source documents and the information entered in the CRF.

## 8.2.2.1. Grading Scales

The grading scales used in this study to assess local reactions and systemic events as described below are derived from the FDA CBER guidelines on toxicity grading scales for healthy adult volunteers enrolled in preventive vaccine clinical trials.<sup>12</sup>

#### 8.2.2.2. Local Reactions

During the reactogenicity e-diary reporting period, participants will be asked to assess redness, swelling, and pain at the injection site and to record the symptoms in the reactogenicity e-diary. If a local reaction persists beyond the end of the reactogenicity e-diary period following vaccination, the participant will be requested to report that information. The investigator will enter this additional information in the CRF.

Redness and swelling will be measured and recorded in measuring device units (range: 1 to 21) and then categorized during analysis as absent, mild, moderate, or severe based on the grading scale in Table 1. Measuring device units can be converted to centimeters according to the following formula: 1 measuring device unit = 0.5 cm. Pain at the injection site will be assessed by the participant as absent, mild, moderate, or severe according to the grading scale in Table 1.

If a Grade 3 local reaction is reported in the reactogenicity e-diary, a telephone contact should occur to ascertain further details and determine whether a site visit is clinically indicated. Only an investigator or medically qualified person is able to classify a participant's local reaction as Grade 4. If a participant experiences a confirmed Grade 4 local reaction, the investigator must immediately notify the sponsor and, if it is determined to be related to the administration of the study intervention, further vaccinations will be discontinued in that participant.

**Table 1. Local Reaction Grading Scale** 

| | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Pain at the injection site | Does not interfere with activity | Interferes with activity | Prevents daily activity | Emergency room visit<br>or hospitalization for<br>severe pain |
| Redness | >2.0 cm to 5.0 cm<br>(5 to 10 measuring<br>device units) | >5.0 cm to 10.0 cm<br>(11 to 20 measuring<br>device units) | >10 cm<br>(≥21 measuring<br>device units) | Necrosis or exfoliative dermatitis |
| Swelling | >2.0 cm to 5.0 cm<br>(5 to 10 measuring<br>device units) | >5.0 cm to 10.0 cm<br>(11 to 20 measuring<br>device units) | >10 cm<br>(≥21 measuring<br>device units) | Necrosis |

## 8.2.2.3. Systemic Events

During the reactogenicity e-diary reporting period, participants will be asked to assess vomiting, diarrhea, headache, fatigue, chills, new or worsened muscle pain, and new or worsened joint pain and to record the symptoms in the reactogenicity e-diary. The symptoms will be assessed by the participant as absent, mild, moderate, or severe according to the grading scale in Table 2.

If a Grade 3 systemic event is reported in the reactogenicity e-diary, a telephone contact should occur to ascertain further details and determine whether a site visit is clinically indicated. Only an investigator or medically qualified person is able to classify a participant's systemic event as Grade 4. If a participant experiences a confirmed Grade 4 systemic event, the investigator must immediately notify the sponsor and, if it is determined to be related to the administration of the study intervention, further vaccinations will be discontinued in that participant.

**Table 2.** Systemic Event Grading Scale

| | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Vomiting | 1-2 times in<br>24 hours | >2 times in 24 hours | Requires IV<br>hydration | Emergency room visit<br>or hospitalization for<br>hypotensive shock |
| Diarrhea | 2 to 3 loose stools in 24 hours | 4 to 5 loose stools in 24 hours | 6 or more loose stools<br>in 24 hours | Emergency room visit or hospitalization for severe diarrhea |
| Headache | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe headache |
| Fatigue/tiredness | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe fatigue |
| Chills | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe chills |
| New or worsened<br>muscle pain | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit<br>or hospitalization for<br>severe new or worsened<br>muscle pain |
| New or worsened joint pain | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit<br>or hospitalization for<br>severe new or worsened<br>joint pain |

Abbreviation: IV = intravenous.

During the 7 days following each vaccination, potential COVID-19 symptoms that overlap with solicited systemic events (ie, fever, chills, new or increased muscle pain, diarrhea, vomiting) should be assessed by the investigator.

If, in the investigator's opinion, the symptoms are considered more likely to be vaccine reactogenicity, but a participant is required to demonstrate that he or she is SARS-CoV-2—negative, a local SARS-CoV-2 test may be performed: if positive, the symptoms should be recorded as an AE rather than as systemic events in the reactogenicity e-diary.

#### 8.2.2.4. Fever

In order to record information on fever, a thermometer will be given to participants with instructions on how to measure oral temperature at home. Temperature will be collected in the reactogenicity e-diary in the evening daily during the reactogenicity e-diary reporting period. It will also be collected at any time during the reactogenicity e-diary data collection periods when fever is suspected. Fever is defined as an oral temperature ≥38.0°C (100.4°F). The highest temperature for each day will be recorded in the reactogenicity e-diary. Temperature will be measured and recorded to 1 decimal place. Temperatures recorded in degrees Fahrenheit will be programmatically converted to degrees Celsius and then categorized according to the scale shown in Table 3 during analysis.

If a fever of ≥39.0°C (102.1°F) is reported in the reactogenicity e-diary, a telephone contact should occur to ascertain further details and determine whether a site visit is clinically indicated. Only an investigator or medically qualified person is able to confirm a participant's fever as >40.0°C (>104.0°F). If a participant experiences a confirmed fever >40.0°C (>104.0°F), the investigator must immediately notify the sponsor and, if it is determined to be related to the administration of the study intervention, further vaccinations will be discontinued in that participant.

Table 3. Scale for Fever

| ≥38.0-38.4°C (100.4-101.1°F) |
|------------------------------|
| >38.4-38.9°C (101.2-102.0°F) |
| >38.9-40.0°C (102.1-104.0°F) |
| >40.0°C (>104.0°F) |

## 8.2.2.5. Antipyretic Medication

The use of antipyretic medication to treat symptoms associated with study intervention administration will be recorded in the reactogenicity e-diary daily during the reporting period (Day 1 through Day 7).

#### **8.2.3. Pregnancy Testing**

Pregnancy tests may be urine or serum tests, but must have a sensitivity of at least 25 mIU/mL. Pregnancy tests will be performed in WOCBP at the times listed in the SoA, immediately before the administration of each vaccine dose. A negative pregnancy test result will be required prior to the participant's receiving the study intervention. Pregnancy tests

may also be repeated if requested by IRBs/ECs or if required by local regulations. In the case of a positive confirmed pregnancy, the participant will be withdrawn from administration of study intervention but may remain in the study.

#### 8.3. Adverse Events and Serious Adverse Events

The definitions of an AE and an SAE can be found in Appendix 3.

AEs will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).

The investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and remain responsible to pursue and obtain adequate information both to determine the outcome and to assess whether the event meets the criteria for classification as an SAE or caused the participant to discontinue the study intervention (see Section 7.1).

Each participant will be questioned about the occurrence of AEs in a nonleading manner.

In addition, the investigator may be requested by Pfizer Safety to obtain specific follow-up information in an expedited fashion.

## 8.3.1. Time Period and Frequency for Collecting AE and SAE Information

The time period for actively eliciting and collecting AEs and SAEs ("active collection period") for each participant begins from the time the participant provides informed consent, which is obtained before the participant's participation in the study (ie, before undergoing any study-related procedure and/or receiving study intervention), through and including Visit 3 (1-month follow-up). In addition, any AEs occurring up to 48 hours after the blood draw and nasal swab collection at Visit 3 reported by the participant must be recorded in the CRF. SAEs will be collected from the time the participant provides informed consent through approximately 1 month after the last dose of study intervention (Visit 3).

For all participants receiving Dose 3, AEs and SAEs will be collected from the time the participant provides informed consent for the receipt of Dose 3 at Visit 101 through Visit 102.

Follow-up by the investigator continues throughout and after the active collection period and until the AE or SAE or its sequelae resolve or stabilize at a level acceptable to the investigator and Pfizer concurs with that assessment.

For participants who are screen failures, the active collection period ends when screen failure status is determined.

If the participant withdraws from the study and also withdraws consent for the collection of future information, the active collection period ends when consent is withdrawn.

If a participant definitively discontinues or temporarily discontinues study intervention because of an AE or SAE, the AE or SAE must be recorded on the CRF and the SAE reported using the Vaccine SAE Reporting Form.

Investigators are not obligated to actively seek AEs or SAEs after the participant has concluded study participation. However, if the investigator learns of any SAE, including a death, at any time after a participant has completed the study, and he/she considers the event to be reasonably related to the study intervention, the investigator must promptly report the SAE to Pfizer using the Vaccine SAE Reporting Form.

## 8.3.1.1. Reporting SAEs to Pfizer Safety

All SAEs occurring in a participant during the active collection period as described in Section 8.3.1 are reported to Pfizer Safety on the Vaccine SAE Reporting Form immediately upon awareness and under no circumstance should this exceed 24 hours, as indicated in Appendix 3. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.

## 8.3.1.2. Recording Nonserious AEs and SAEs on the CRF

All nonserious AEs and SAEs occurring in a participant during the active collection period, which begins after obtaining informed consent as described in Section 8.3.1, will be recorded on the AE section of the CRF.

The investigator is to record on the CRF all directly observed and all spontaneously reported AEs and SAEs reported by the participant.

#### 8.3.2. Method of Detecting AEs and SAEs

The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Section 10.3.

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and nonleading verbal questioning of the participant is the preferred method to inquire about AE occurrences.

#### 8.3.3. Follow-up of AEs and SAEs

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. For each event, the investigator must pursue and obtain adequate information until resolution, stabilization, the event is otherwise explained, or the participant is lost to follow-up (as defined in Section 7.3).

In general, follow-up information will include a description of the event in sufficient detail to allow for a complete medical assessment of the case and independent determination of possible causality. Any information relevant to the event, such as concomitant medications and illnesses, must be provided. In the case of a participant death, a summary of available autopsy findings must be submitted as soon as possible to Pfizer Safety.

Further information on follow-up procedures is given in Appendix 3.

## 8.3.4. Regulatory Reporting Requirements for SAEs

Prompt notification by the investigator to the sponsor of an SAE is essential so that legal obligations and ethical responsibilities towards the safety of participants and the safety of a study intervention under clinical investigation are met.

The sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study intervention under clinical investigation. The sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, IRBs/ECs, and investigators.

Investigator safety reports must be prepared for SUSARs according to local regulatory requirements and sponsor policy and forwarded to investigators as necessary.

An investigator who receives SUSARs or other specific safety information (eg, summary or listing of SAEs) from the sponsor will review and then file it along with the SRSD(s) for the study and will notify the IRB/EC, if appropriate according to local requirements.

## 8.3.5. Exposure During Pregnancy or Breastfeeding, and Occupational Exposure

Exposure to the study intervention under study during pregnancy or breastfeeding and occupational exposure are reportable to Pfizer Safety within 24 hours of investigator awareness.

## **8.3.5.1.** Exposure During Pregnancy

An EDP occurs if:

- A female participant is found to be pregnant while receiving or after discontinuing study intervention.
- A male participant who is receiving or has discontinued study intervention exposes a female partner prior to or around the time of conception.
- A female is found to be pregnant while being exposed or having been exposed to study intervention due to environmental exposure. Below are examples of environmental exposure during pregnancy:
  - A female family member or healthcare provider reports that she is pregnant after having been exposed to the study intervention by inhalation or skin contact.
  - A male family member or healthcare provider who has been exposed to the study intervention by inhalation or skin contact then exposes his female partner prior to or around the time of conception.

The investigator must report EDP to Pfizer Safety within 24 hours of the investigator's awareness, irrespective of whether an SAE has occurred. The initial information submitted PFIZER CONFIDENTIAL

should include the anticipated date of delivery (see below for information related to termination of pregnancy).

- If EDP occurs in a participant or a participant's partner, the investigator must report this information to Pfizer Safety on the Vaccine SAE Reporting Form and an EDP Supplemental Form, regardless of whether an SAE has occurred. Details of the pregnancy will be collected after the start of study intervention and until 1 month after the last dose of study intervention.
- If EDP occurs in the setting of environmental exposure, the investigator must report information to Pfizer Safety using the Vaccine SAE Reporting Form and EDP Supplemental Form. Since the exposure information does not pertain to the participant enrolled in the study, the information is not recorded on a CRF; however, a copy of the completed Vaccine SAE Reporting Form is maintained in the ISF.

Follow-up is conducted to obtain general information on the pregnancy and its outcome for all EDP reports with an unknown outcome. The investigator will follow the pregnancy until completion (or until pregnancy termination) and notify Pfizer Safety of the outcome as a follow-up to the initial EDP Supplemental Form. In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless preprocedure test findings are conclusive for a congenital anomaly and the findings are reported).

Abnormal pregnancy outcomes are considered SAEs. If the outcome of the pregnancy meets the criteria for an SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly), the investigator should follow the procedures for reporting SAEs. Additional information about pregnancy outcomes that are reported to Pfizer Safety as SAEs follows:

- Spontaneous abortion including miscarriage and missed abortion;
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as SAEs when the investigator assesses the infant death as related or possibly related to exposure to the study intervention.

Additional information regarding the EDP may be requested by the sponsor. Further follow-up of birth outcomes will be handled on a case-by-case basis (eg, follow-up on preterm infants to identify developmental delays). In the case of paternal exposure, the investigator will provide the participant with the Pregnant Partner Release of Information Form to deliver to his partner. The investigator must document in the source documents that the participant was given the Pregnant Partner Release of Information Form to provide to his partner.

## 8.3.5.2. Exposure During Breastfeeding

An exposure during breastfeeding occurs if:

- A female participant is found to be breastfeeding while receiving or after discontinuing study intervention.
- A female is found to be breastfeeding while being exposed or having been exposed to study intervention (ie, environmental exposure). An example of environmental exposure during breastfeeding is a female family member or healthcare provider who reports that she is breastfeeding after having been exposed to the study intervention by inhalation or skin contact.

The investigator must report exposure during breastfeeding to Pfizer Safety within 24 hours of the investigator's awareness, irrespective of whether an SAE has occurred. The information must be reported using the Vaccine SAE Reporting Form. When exposure during breastfeeding occurs in the setting of environmental exposure, the exposure information does not pertain to the participant enrolled in the study, so the information is not recorded on a CRF. However, a copy of the completed Vaccine SAE Reporting Form is maintained in the ISF.

An exposure during breastfeeding report is not created when a Pfizer drug specifically approved for use in breastfeeding women (eg, vitamins) is administered in accord with authorized use. However, if the infant experiences an SAE associated with such a drug, the SAE is reported together with the exposure during breastfeeding.

## 8.3.5.3. Occupational Exposure

An occupational exposure occurs when a person receives unplanned direct contact with the study intervention, which may or may not lead to the occurrence of an AE. Such persons may include healthcare providers, family members, and other roles that are involved in the trial participant's care.

The investigator must report occupational exposure to Pfizer Safety within 24 hours of the investigator's awareness, regardless of whether there is an associated SAE. The information must be reported using the Vaccine SAE Reporting Form. Since the information does not pertain to a participant enrolled in the study, the information is not recorded on a CRF; however, a copy of the completed Vaccine SAE Reporting Form is maintained in the ISF.

#### 8.3.6. Cardiovascular and Death Events

Not applicable.

## 8.3.7. Disease-Related Events and/or Disease-Related Outcomes Not Qualifying as AEs or SAEs

Not applicable.

## 8.3.8. Adverse Events of Special Interest

This section provides information on AESIs that may be detected during the study:

- Confirmed COVID-19 diagnosis (clinical signs/symptoms and positive SARS-CoV-2 NAAT test)
- A confirmed diagnosis of myocarditis or pericarditis. See Section 8.13 for additional procedures for monitoring of potential myocarditis or pericarditis.

All AESIs must be reported as an AE or SAE following the procedures described in Section 8.3.1 through Section 8.3.4. An AESI is to be recorded as an AE or SAE on the CRF. In addition, an AESI that is also an SAE must be reported using the Vaccine SAE Reporting Form.

## 8.3.8.1. Lack of Efficacy

Lack of efficacy is reportable to Pfizer Safety only if associated with an SAE.

#### 8.3.9. Medical Device Deficiencies

Not applicable.

#### 8.3.10. Medication Errors

Medication errors may result from the administration or consumption of the study intervention by the wrong participant, or at the wrong time, or at the wrong dosage strength.

Exposures to the study intervention under study may occur in clinical trial settings, such as medication errors.

| Safety Event | Recorded on the CRF | Reported on the Vaccine SAE Reporting Form to Pfizer Safety Within 24 Hours of Awareness |
|---|---|---|
| Medication errors | All (regardless of whether associated with an AE) | Only if associated with an SAE |

#### Medication errors include:

- Medication errors involving participant exposure to the study intervention;
- Potential medication errors or uses outside of what is foreseen in the protocol that do or do not involve the study participant;
- The administration of expired study intervention;
- The administration of an incorrect study intervention;
- The administration of an incorrect dosage;

• The administration of study intervention that has undergone temperature excursion from the specified storage range, unless it is determined by the sponsor that the study intervention under question is acceptable for use.

Such medication errors occurring to a study participant are to be captured on the medication error page of the CRF, which is a specific version of the AE page.

In the event of a medication dosing error, the sponsor should be notified within 24 hours.

Whether or not the medication error is accompanied by an AE, as determined by the investigator, the medication error is recorded on the medication error page of the CRF and, if applicable, any associated AE(s), serious and nonserious, are recorded on the AE page of the CRF.

Medication errors should be reported to Pfizer Safety within 24 hours on a Vaccine SAE Reporting Form **only when associated with an SAE**.

#### 8.4. Treatment of Overdose

For this study, any dose of study intervention greater than 1 dose of study intervention within a 24-hour time period will be considered an overdose.

Pfizer does not recommend specific treatment for an overdose.

In the event of an overdose, the investigator should:

- 1. Contact the medical monitor within 24 hours.
- 2. Closely monitor the participant for any AEs/SAEs.
- 3. Document the quantity of the excess dose as well as the duration of the overdose in the CRF.
- 4. Overdose is reportable to Safety only when associated with an SAE.

Decisions regarding dose interruptions or modifications will be made by the investigator in consultation with the medical monitor based on the clinical evaluation of the participant.

#### 8.5. Pharmacokinetics

Pharmacokinetic parameters are not evaluated in this study.

#### 8.6. Pharmacodynamics

Pharmacodynamic parameters are not evaluated in this study.

#### 8.7. Genetics

Genetics (specified analyses) are not evaluated in this study.

## 8.8. Biomarkers

Biomarkers are not evaluated in this study.

## 8.9. Immunogenicity Assessments

Immunogenicity assessments are described in Section 8.1.

#### 8.10. Health Economics

Health economics/medical resource utilization and health economics parameters are not evaluated in this study.

## 8.11. Study Procedures

## **8.11.1.** Visit 1 – Vaccination 1 (Day 1)

Before enrollment and before any study-related procedures are performed, voluntary, written, study-specific informed consent will be obtained from the participant. Each signature on the ICD must be personally dated by the signatory. The investigator or his or her designee will also sign the ICD. A copy of the signed and dated ICD must be given to the participant. The source data must reflect that the informed consent was obtained before participation in the study.

It is anticipated that the procedures below will be conducted in a stepwise manner. The visit may be conducted across 2 consecutive days; if so, all steps from assessing the inclusion and exclusion criteria onward must be conducted on the same day.

- Assign a single participant number using the IRT system.
- Obtain the participant's demography (including date of birth, sex, race, and ethnicity). The full date of birth will be collected to critically evaluate the immune response and safety profile by age.
- Obtain any medical history of clinical significance.
- Perform a clinical assessment. If the clinical assessment indicates that a physical examination is necessary to comprehensively evaluate the participant, perform a physical examination and record any findings in the source documents and, if clinically significant, record on the medical history CRF.
- Measure the participant's height and weight.
- Ensure and document that all of the inclusion criteria and none of the exclusion criteria are met.
- Measure the participant's body temperature.
- Perform urine pregnancy test on WOCBP as described in Section 8.2.3.

- Discuss contraceptive use as described in Section 5.3.1.
- Record nonstudy vaccinations as described in Section 6.5.
- Collect a blood sample of approximately 20 mL for immunogenicity testing and to test for prior COVID-19. Please refer to the ISF for further instructions.
- Obtain a nasal (midturbinate) swab (collected by site staff) for determination of current SARS-CoV-2 status. Please refer to the ISF for further instructions.
- A blinded site staff member obtains the randomization number using the IRT system. An unblinded site staff member then enters the participant number (SSID) and randomization number to assign the study intervention allocation number.
- Unblinded site staff member(s) will dispense/administer 1 dose of study intervention into the deltoid muscle of the (preferably) nondominant arm. Please refer to the IP manual for further instruction on this process.
- Blinded site staff must observe the participant for at least 30 minutes after study intervention administration for any acute reactions. Record any acute reactions (including time of onset) in the participant's source documents and on the AE page of the CRF, and on an SAE form as applicable.
- Explain the e-diary technologies available for this study (Section 8.2.2), and assist the participant in downloading the study application onto the participant's own device or issue a provisioned device if required.
  - Provide instructions on reactogenicity e-diary completion and ask the participant to complete the reactogenicity e-diary from Day 1 through Day 7, with Day 1 being the day of vaccination.
- Ask the participant to contact the site staff or investigator immediately if the participant experiences any of the following from Day 1 through Day 7 after vaccination (where Day 1 is the day of vaccination) to determine if an unscheduled reactogenicity visit is required:
  - Fever >39.0°C (>102.1°F).
  - Redness or swelling at the injection site measuring greater than 10 cm (>20 measuring device units).
  - Severe pain at the injection site.
  - Any severe systemic event.
- Issue a measuring device to measure local reactions at the injection site and a thermometer for recording daily temperatures and provide instructions on their use.


- Record AEs/SAEs as described in Section 8.3.
- Ask the participant to contact the site staff or investigator if a medically attended event (eg, doctor's visit, emergency room visit) or hospitalization occurs.
- Ask the participant to contact the site staff or investigator if he/she develops symptoms of a COVID-19 infection, as defined by the CDC, <sup>13</sup> including:
  - New or increased cough;
  - New or increased shortness of breath;
  - Chills;
  - New or increased muscle pain;
  - New loss of taste/smell;
  - Sore throat;
  - Diarrhea;
  - Vomiting.
- Schedule an appointment for the participant to return for the next study visit.
- Remind the participant to bring the reactogenicity e-diary to the next visit.
- Complete the source documents.
- The investigator or an authorized designee completes the CRFs and an unblinded dispenser/administrator updates the study intervention accountability records.

The investigator or appropriately qualified designee reviews the reactogenicity e-diary data online following vaccination to evaluate participant compliance and as part of the ongoing safety review. Daily review is optimal during the active diary period.

## 8.11.2. Visit 2 – Vaccination 2 (19 to 23 Days After Visit 1)

- Record AEs/SAEs as described in Section 8.3.
- Review the participant's reactogenicity e-diary data. Collect stop dates of any reactogenicity e-diary events ongoing on the last day that the reactogenicity e-diary was completed and record stop dates in the CRF if required.
- Perform urine pregnancy test on WOCBP as described in Section 8.2.3.

- Discuss contraceptive use as described in Section 5.3.1.
- Record nonstudy vaccinations as described in Section 6.5.
- Record details of any of the prohibited medications specified in Section 6.5.1 received by the participant if required for his or her clinical care.
- Ensure and document that all of the inclusion criteria and none of the exclusion criteria are met. If these eligibility criteria are not met, the participant may not receive further study intervention but will remain in the study to be evaluated for safety, immunogenicity, and efficacy (see Section 7).
  - A positive SARS-CoV-2 NAAT result without symptoms or a COVID-19 diagnosis (signs/symptoms only or signs/symptoms and a positive SARS-CoV-2 NAAT result) should not result in discontinuation of study intervention.
  - If study intervention (Dose 2) has been delayed per the criteria for temporary delay, because of febrile or other acute illness (Item 1, criteria for temporary delay), and the investigator later diagnoses the signs and symptoms as COVID-19 (with or without a positive SARS-CoV-2 NAAT result), the participant should not be discontinued from any further doses of study intervention.
- Measure the participant's body temperature.
- Ensure that the participant meets none of the temporary delay criteria as described in Section 5.5.
- Unblinded site staff member(s) will dispense/administer 1 dose of study intervention into the deltoid muscle of the (preferably) nondominant arm. Please refer to the IP manual for further instruction on this process.
- Blinded site staff must observe the participant for at least 30 minutes after study intervention administration for any acute reactions. Record any acute reactions (including time of onset) in the participant's source documents and on the AE page of the CRF, and on an SAE form as applicable.
- Ensure the participant has a measuring device to measure local reactions at the injection site and a thermometer for recording daily temperatures.
- Ensure the participant remains comfortable with the chosen e-diary platform, confirm instructions on e-diary completion, and ask the participant to complete the reactogenicity e-diary from Day 1 through Day 7, with Day 1 being the day of vaccination.
- Ask the participant to contact the site staff or investigator immediately if the participant experiences any of the following from Day 1 through Day 7 after

vaccination (where Day 1 is the day of vaccination) to determine if an unscheduled reactogenicity visit is required:

- Fever  $\ge 39.0^{\circ}\text{C} (\ge 102.1^{\circ}\text{F})$ .
- Redness or swelling at the injection site measuring greater than 10 cm (>20 measuring device units).
- Severe pain at the injection site.
- Any severe systemic event.
- Ask the participant to contact the site staff or investigator if a medically attended event (eg, doctor's visit, emergency room visit) or hospitalization occurs.
- Ask the participant to contact the site staff or investigator if he/she develops symptoms of a COVID-19 infection, as defined by the CDC, <sup>13</sup> including:
  - New or increased cough;
  - New or increased shortness of breath;
  - Chills:
  - New or increased muscle pain;
  - New loss of taste/smell;
  - Sore throat;
  - Diarrhea;
  - Vomiting.
- Schedule an appointment for the participant to return for the next study visit.
- Remind the participant to bring the reactogenicity e-diary to the next visit.
- Complete the source documents.
- The investigator or an authorized designee completes the CRFs and an unblinded dispenser/administrator updates the study intervention accountability records.

The investigator or appropriately qualified designee reviews the reactogenicity e-diary data online following vaccination to evaluate participant compliance and as part of the ongoing safety review. Daily review is optimal during the active diary period.

## 8.11.3. Visit 3 – 1-Month Follow-up (28 to 35 Days After Visit 2)

- Record AEs/SAEs as described in Section 8.3.
- Review the participant's reactogenicity e-diary data. Collect stop dates of any reactogenicity e-diary events ongoing on the last day that the reactogenicity e-diary was completed and record stop dates in the CRF if required.
- Record nonstudy vaccinations as described in Section 6.5.
- Record details of any of the prohibited medications specified in Section 6.5.1 received by the participant if required for his or her clinical care.
- Discuss contraceptive use as described in Section 5.3.1.
- Collect a blood sample of approximately 20 mL for immunogenicity testing and to test for prior COVID-19.
- Obtain a nasal (midturbinate) swab (collected by site staff) for determination of current SARS-CoV-2 status.
- Collect the participant's reactogenicity e-diary or assist the participant to remove the study application from his or her own personal device.
- Complete the source documents.
- The investigator or an authorized designee completes the CRFs.

#### 8.11.4. Unscheduled Visits for a Grade 3 or Suspected Grade 4 Reaction

If a Grade 3 local reaction (Section 8.2.2.2), systemic event (Section 8.2.2.3), or fever (Section 8.2.2.4) is reported in the reactogenicity e-diary, a telephone contact should occur to ascertain further details and determine whether a site visit is clinically indicated. If a suspected Grade 4 local reaction (Section 8.2.2.2), systemic event (Section 8.2.2.3), or fever (Section 8.2.2.4) is reported in the reactogenicity e-diary, a telephone contact or site visit should occur to confirm whether the event meets the criteria for Grade 4.

A site visit must be scheduled as soon as possible to assess the participant unless any of the following is true:

- The participant is unable to attend the unscheduled visit.
- The local reaction/systemic event is no longer present at the time of the telephone contact.
- The participant recorded an incorrect value in the reactogenicity e-diary (confirmation of a reactogenicity e-diary data entry error).

• The PI or authorized designee determined it was not needed.

This telephone contact will be recorded in the participant's source documentation and the CRF.

If the participant is unable to attend the unscheduled visit, or the PI or authorized designee determined it was not needed, any ongoing local reactions/systemic events must be assessed at the next study visit.

During the unscheduled visit, the reactions should be assessed by the investigator or a medically qualified member of the study staff such as a study physician or a study nurse, as applicable to the investigator's local practice, who will:

- Measure body temperature (°F/°C).
- Measure minimum and maximum diameters of redness (if present).
- Measure minimum and maximum diameters of swelling (if present).
- Assess injection site pain (if present) in accordance with the grades provided in Section 8.2.2.2.
- Assess systemic events (if present) in accordance with the grades provided in Section 8.2.2.3.
- Assess for other findings associated with the reaction and record on the AE page of the CRF, if appropriate.

The investigator or an authorized designee will complete the unscheduled visit assessment page of the CRF.

# 8.12. Study Procedures for Participants Who Accept the Offer to Receive Dose 38.12.1. Visit 101 – Vaccination 3 (At Least 90 Days After Visit 2)

Before Vaccination 3 and before any study-related procedures are performed, voluntary, written, study-specific informed consent will be obtained from the participant. Each signature on the ICD must be personally dated by the signatory. The investigator or his or her designee will also sign the ICD. A copy of the signed and dated ICD must be given to the participant. The source data must reflect that the informed consent was obtained before participation in the study.

It is anticipated that the procedures below will be conducted in a stepwise manner.

- Confirm that the participant originally received lyophilized formulation of BNT162b2 at Vaccinations 1 and 2. Secondary confirmation by another site staff is required.
- Measure the participant's body temperature.

- Perform urine pregnancy test on WOCBP as described in Section 8.2.3.
- Discuss contraceptive use as described in Section 5.3.1.
- Record nonstudy vaccinations as described in Section 6.5.
- Record details of any of the prohibited medications specified in Section 6.5.1 received by participant if required for his or her clinical care.
- Review and consider inclusion criteria 2, 3, 4, and 5 and exclusion criteria.
- Confirm that the participant meets all of the inclusion criteria and does not meet exclusion criteria 1, 3, 5, 6, 7, 10, 11, 12, 13, and 14.
- Ensure that the participant does not meet any of the temporary delay criteria as described in Section 5.5.
- Collect a blood sample of approximately 20 mL for immunogenicity testing. Please refer to the ISF for further instructions.
- Obtain a nasal (midturbinate) swab (collected by site staff) for determination of current SARS-CoV-2 status. Please refer to the ISF for further instructions.
- Obtain the participant's vaccine allocation vial using the IRT system.
- Dispense/administer 1 dose of study intervention into the deltoid muscle of the (preferably) nondominant arm. Please refer to the IP manual for further instruction on this process.
- Observe the participant for at least 30 minutes after study intervention administration for any acute reactions. Record any acute reactions (including time of onset) in the participant's source documents and on the AE page of the CRF, and on an SAE form as applicable.
- Issue a measuring device to measure local reactions at the injection site and a thermometer for recording daily temperatures and provide instructions on their use.
- Remind the participant of the e-diary technologies available for this study (Section 8.2.2), and assist the participant in downloading the study application onto the participant's own device or issue a provisioned device if required.
  - Provide instructions on reactogenicity e-diary completion and ask the participant to complete the reactogenicity e-diary from Day 1 through Day 7, with Day 1 being the day of vaccination.

- Ask the participant to contact the site staff or investigator immediately if the participant experiences any of the following from Day 1 through Day 7 after vaccination (where Day 1 is the day of vaccination) to determine if an unscheduled reactogenicity visit is required:
  - Fever  $\ge 39.0^{\circ}\text{C} (\ge 102.1^{\circ}\text{F})$ .
  - Redness or swelling at the injection site measuring greater than 10 cm (>20 measuring device units).
  - Severe pain at the injection site.
  - Any severe systemic event.
- Record AEs/SAEs as described in Section 8.3.
- Ask the participant to contact the site staff or investigator if a medically attended event (eg, doctor's visit, emergency room visit) or hospitalization occurs.
- Ask the participant to contact the site staff or investigator if he/she develops symptoms of a COVID-19 infection, as defined by the CDC, <sup>13</sup> including:
  - New or increased cough;
  - New or increased shortness of breath;
  - Chills;
  - New or increased muscle pain;
  - New loss of taste/smell;
  - Sore throat;
  - Diarrhea;
  - Vomiting.
- Schedule an appointment for the participant to return for the next study visit.
- Remind the participant to bring the reactogenicity e-diary to the next visit.
- Complete the source documents.
- The investigator or an authorized designee completes the CRFs and an unblinded dispenser/administrator updates the study intervention accountability records.

The investigator or appropriately qualified designee reviews the reactogenicity e-diary data online following vaccination to evaluate participant compliance and as part of the ongoing safety review. Daily review is optimal during the active diary period.

## 8.12.2. Visit 102 – 1-Month Follow-up (28 to 35 Days After Visit 101)

- Record AEs/SAEs as described in Section 8.3.
- Review the participant's reactogenicity e-diary data. Collect stop dates of any reactogenicity e-diary events ongoing on the last day that the reactogenicity e-diary was completed and record stop dates in the CRF if required.
- Record nonstudy vaccinations as described in Section 6.5.
- Record details of any of the prohibited medications specified in Section 6.5.1 received by the participant if required for his or her clinical care.
- Discuss contraceptive use as described in Section 5.3.1.
- Collect a blood sample of approximately 20 mL for immunogenicity testing.
- Obtain a nasal (midturbinate) swab (collected by site staff) for determination of current SARS-CoV-2 status. Please refer to the ISF for further instructions.
- Collect the participant's reactogenicity e-diary or assist the participant to remove the study application from his or her own personal device.
- Complete the source documents.
- The investigator or an authorized designee completes the CRFs.

## 8.13. Additional Procedures for Monitoring of Potential Myocarditis or Pericarditis

Any study participant who reports acute chest pain, shortness of breath, palpitations, or any other symptom(s) that might be indicative of myocarditis or pericarditis within 4 weeks of a study vaccination should be specifically evaluated, preferably by a cardiologist, for possible myocarditis or pericarditis.

In addition to a clinical evaluation, the following should be performed:

- ECG
- Troponin level

If myocarditis or pericarditis are suspected based upon the initial evaluation, the following should also be performed:

• Cardiac echocardiogram, and/or

• Cardiac magnetic resonance study

Details of the symptoms reported, and results of the investigations performed, will be recorded in the CRF.

#### 9. STATISTICAL CONSIDERATIONS

Methodology for summary and statistical analyses of the data collected in this study is described here and further detailed in a SAP, which will be maintained by the sponsor. The SAP may modify what is outlined in the protocol where appropriate; however, any major modifications of the primary endpoint definitions or their analyses will also be reflected in a protocol amendment.

## 9.1. Estimands and Statistical Hypotheses

#### 9.1.1. Estimands

The estimands corresponding to each primary and secondary objective are described in the table in Section 3.

The estimands to evaluate the immunogenicity objectives are based on the evaluable immunogenicity population (Section 9.3). These estimands estimate the vaccine effect in the hypothetical settings where participants follow the study schedules and protocol requirements as directed. The estimands address the objective of estimating the maximum potential difference between 2 groups, since the impact of noncompliance is likely to diminish the observed difference between the 2 groups. Missing antibody results will not be imputed. Immunogenicity results that are below the LLOQ will be set to  $0.5 \times LLOQ$  in the analysis; this may be adjusted once additional data on the assay characteristics become available.

In the primary safety objective evaluations, missing reactogenicity e-diary data will not be imputed. Missing AE start dates will be imputed according to Pfizer safety rules. No other missing information will be imputed in the safety analysis.

## 9.1.2. Statistical Hypothesis

The primary immunogenicity objective is to assess the noninferiority of the immune response induced by lyophilized SDV compared to frozen-liquid MDV BNT162b2. The null hypothesis  $(H_0)$  is

$$H_0$$
:  $ln(\mu_1) - ln(\mu_2) \le ln(0.67)$  vs  $H_1$ :  $ln(\mu_1) - ln(\mu_2) > ln(0.67)$ 

where ln(0.67) corresponds to a 1.5-fold margin for noninferiority and

 ln(μ<sub>1</sub>) is the natural log of the geometric mean of full-length S-binding IgG levels measured 1 month after Dose 2 from participants receiving lyophilized SDV BNT162b2;  ln(μ<sub>2</sub>) is the natural log of the geometric mean of full-length S-binding IgG levels measured 1 month after Dose 2 from participants receiving frozen-liquid MDV BNT162b2 control for lyophilized SDV

Noninferiority will be declared if the lower bound of the 2-sided 95% CI for the GMR of lyophilized SDV relative to the corresponding frozen-liquid MDV control is greater than 0.67 (1.5-fold criterion).

#### 9.1.3. Multiplicity Considerations

There is only 1 hypothesis for the primary immunogenicity endpoint, and within-group descriptive summaries will be provided for the secondary immunogenicity endpoint. Consequently, no multiplicity adjustments are applied.

## 9.2. Sample Size Determination

The sample size in Part 1 of the study is based on the noninferiority evaluation for the primary immunogenicity endpoint, full-length S-binding IgG levels 1 month after Dose 2, using a 1.5-fold noninferiority margin for the comparison between lyophilized SDV BNT162b2 relative to frozen-liquid MDV BNT162b2. The second part of the study for assessing the immune responses induced by frozen-liquid BNT162b2 with LNP size at the upper end of specification or RTU BNT162b2 is for descriptive purposes; thus, sample size for this part is not based on statistical considerations.

Common assay standard deviations from each group are assumed to be 0.6456 based on results from Phase 1 of Study C4591001 (BNT162b2 30  $\mu g$ , 18- to 55-year age group). With this standard deviation and the observed GMT difference assumed in the power analysis below, a sample size of 220 evaluable participants per group in Part 1 of the study will provide a power of 90.1% to declare noninferiority of lyophilized BNT162b2 to frozen-liquid MDV for the primary objective (Table 4).

Assuming a nonevaluable rate of 20%, the study will randomize approximately 275 participants to each group in Part 1 of the study to achieve the required number of evaluable participants.

| T 1 1 4 | The state of the s | | • | TA. T • | • • • | A . |
|---|---|---|---|---|---|---|
| Table 4. | POWAR A | lnalveic | tor | Nonin | teriority | Assessment |
| I am T. | | MILALVOIS | 11//1 | 1 44711111 | | |

| Criteria | Standard Deviation<br>(Log Value) <sup>a</sup> | Assumed Observed<br>GMT Difference<br>(Log Scale) | Number of Evaluable<br>Participants per<br>Group | Power <sup>b</sup> |
|---|---|---|---|---|
| Lower limit of 95% CI for GMR (lyophilized SDV | 0.6456 | -0.2 | 220 | 90.1% |
| BNT162b2/frozen-liquid<br>MDV BNT162b2) >0.67 | | | | |

Abbreviations: GMR = geometric mean ratio; GMT = geometric mean titer; MDV = multidose vial; SDV = single-dose vial.

- a. Reference: BNT162b2 (30  $\mu$ g), 18- to 55-year age group (C4591001 Phase 1, N=12). Calculation may be updated if additional information becomes available to better estimate the standard deviation.
- b. At the 0.05 alpha level (2-sided).

## 9.3. Analysis Sets

For purposes of analysis, the following analysis sets are defined:

| Participant Analysis Set | Description |
|---|---|
| Enrolled | All participants who have a signed ICD. |
| Randomized | All participants who are assigned a randomization number in the IWR system. |
| Evaluable immunogenicity | All eligible randomized participants who receive 2 doses of the vaccine to which they are randomized with Dose 2 received within the predefined window, have at least 1 valid and determinate immunogenicity result from the blood sample collected within an appropriate window at 1 month after the Dose 2 visit, are negative for SARS-CoV-2 infection during the study, and have no other important protocol deviations as determined by the clinician. |
| Dose 3 evaluable immunogenicity | All eligible randomized participants who receive 2 doses of lyophilized formulation of BNT162b2 to which they are randomized, with Dose 2 received within the predefined window, receive a third dose of frozen-liquid BNT162b2 formulation, have at least 1 valid and determinate immunogenicity result from the blood sample collected within an appropriate window at the 1-month post–Dose 3 visit, are negative for SARS-CoV-2 infection during the study, and have no other important protocol deviations as determined by the clinician. |
| All-available immunogenicity | All participants who receive at least 1 dose of the study intervention and have at least 1 valid and determinate immunogenicity result after vaccination. |
| Safety | All randomized participants who receive at least 1 dose of the study intervention. |

## 9.4. Statistical Analyses

The SAP will be developed and finalized before any analyses are performed and will describe the analyses and procedures for accounting for missing, unused, and spurious data. This section is a summary of the planned statistical analyses of the primary and secondary endpoints.

#### 9.4.1. General Considerations

Unless stated otherwise, "vaccine group" in this section refers to participants receiving lyophilized SDV, frozen-liquid MDV control for lyophilized SDV, frozen-liquid BNT162b2 with LNP size at the upper end of specification, or RTU BNT162b2. CIs for all endpoints in

the statistical analysis will be presented as 2-sided at the 95% level unless specified otherwise.

For all the immunogenicity endpoints, the analysis will be based on the evaluable immunogenicity population or Dose 3 evaluable immunogenicity population. An additional analysis will be performed based on the all-available immunogenicity population if there is a large enough difference in sample size between the all-available immunogenicity population and the evaluable immunogenicity population. Participants will be summarized according to the vaccine group to which they were randomized.

The safety analyses will be based on the safety population. Participants will be summarized by vaccine group according to the study interventions they actually received.

## 9.4.1.1. Analysis for Binary Data

Descriptive statistics for categorical variables (eg, proportions) are the percentage (%), the numerator (n) and the denominator (N) used in the percentage calculation, and the 95% CIs where applicable.

The exact 95% CI for binary endpoints for each group will be computed using the F distribution (Clopper-Pearson).

#### 9.4.1.2. Analysis for Continuous Data

Unless otherwise stated, descriptive statistics for continuous variables are n, mean, median, standard deviation, minimum, and maximum.

#### 9.4.1.2.1. Geometric Mean Ratios

The GMRs will be calculated as the mean of the difference of logarithmically transformed assay results between 2 vaccine groups and exponentiating the mean. Two-sided CIs will be obtained by calculating CIs using Student's t-distribution for the mean difference of the logarithmically transformed assay results and exponentiating the confidence limits.

## 9.4.1.2.2. Geometric Means

The geometric means will be calculated as the mean of the assay results after making the logarithmic transformation and then exponentiating the mean to express results on the original scale. Two-sided 95% CIs will be obtained by taking log transforms of assay results, calculating the 95% CI with reference to Student's t-distribution, and then exponentiating the confidence limits.

#### 9.4.1.2.3. Geometric Mean Fold Rises

GMFRs are defined as ratios of the results after vaccination to the results before vaccination. GMFRs are limited to participants with nonmissing values at both time points.

GMFRs will be calculated as the mean of the difference of logarithmically transformed assay results (later time point minus earlier time point) and exponentiating the mean. The associated 2-sided 95% CIs will be obtained by constructing CIs using Student's


t-distribution for the mean difference on the logarithm scale and exponentiating the confidence limits.

## 9.4.1.2.4. Reverse Cumulative Distribution Curve

Empirical RCDCs will plot proportions of participants with values equal to or exceeding a specified assay value versus the indicated assay value, for all observed assay values. Data points will be joined by a step function with data points on the left side of the step.

## 9.4.2. Primary Endpoint(s)

| Endpoint | Statistical Analysis Methods |
|---|---|
| Immunogenicity | GMR of full-length S-binding IgG levels in participants receiving lyophilized SDV BNT162b2 compared to frozen-liquid MDV BNT162b2 control for lyophilized SDV |
| | For full-length S-binding IgG levels, the GMR at 1 month after Dose 2 will be provided along with associated 2-sided 95% CIs (see Section 9.4.1.2.1). |
| | Noninferiority will be declared if the lower limit of the 2-sided 95% CI for the GMR is greater than 0.67. |
| Safety | Descriptive statistics will be provided for each reactogenicity endpoint for each dose and vaccine group. Local reactions and systemic events from Day 1 through Day 7 after each vaccination (where Day 1 is the day of vaccination) will be presented by severity and cumulatively across severity levels. Descriptive summary statistics will include counts and percentages of participants with the indicated endpoint and the associated Clopper-Pearson 95% CIs (see Section 9.4.1.1). |
| | AEs and SAEs will be categorized according to MedDRA terms. Counts, percentages, and the associated Clopper-Pearson 95% CIs of AEs and SAEs from Dose 1 through 1 month after Dose 2 will be provided for each vaccine group. |

## 9.4.3. Secondary Endpoint(s)

| Endpoint | Statistical Analysis Methods |
|---|---|
| Immunogenicity | GMCs of full-length S-binding IgG levels |
| | For full-length S-binding IgG levels, GMCs and 2-sided 95% CIs will be provided for each vaccine group in Part 1 of the study (lyophilized BNT162b2 in SDVs and frozen-liquid BNT162b2 in MDVs) at baseline (before Dose 1) and at 1 month after Dose 2. |
| | Statistical methods are described in Section 9.4.1.2.2. |
| | GMFRs of full-length S-binding IgG levels |
| | For full-length S-binding IgG levels, the GMFRs and 2-sided 95% CIs will be provided for each vaccine group in Part 1 of the study (lyophilized BNT162b2 in SDVs and frozen-liquid BNT162b2 in MDVs) from baseline (before Dose 1) to 1 month after Dose 2. |


| Endpoint | Statistical Analysis Methods |
|---|---|
| | GMFRs will be limited to participants with nonmissing values prior to the first dose and at the postvaccination time point. The statistical methods are described in Section 9.4.1.2.3. |

## 9.4.4. Exploratory Endpoint(s)

| Endpoint | Statistical Analysis Methods |
|---|---|
| Safety | Descriptive statistics will be provided for each reactogenicity endpoint in participants who originally received 2 doses of lyophilized formulation of BNT162b2 and received frozen-liquid BNT162b2 formulation as a third dose. Local reactions and systemic events from Day 1 through Day 7 after the third dose (where Day 1 is the day of the third dose) will be presented by severity and cumulatively across severity levels. Descriptive summary statistics will include counts and percentages of participants with the indicated endpoint and the associated Clopper-Pearson 95% CIs (see Section 9.4.1.1). |
| | AEs and SAEs will be categorized according to MedDRA terms. Counts and percentages of participants with AEs and SAEs from Dose 3 through 1 month after Dose 3 will be provided, along with the associated Clopper-Pearson 95% CIs. |
| Immunogenicity | GMR of frozen-liquid BNT162b2 with LNP size at the upper end of specification relative to frozen-liquid BNT162b2 in MDVs at 1 month after Dose 2 |
| | For full-length S-binding IgG levels and/or SARS-CoV-2 neutralizing titers, the GMR at 1 month after Dose 2 will be provided along with associated 2-sided 95% CIs (see Section 9.4.1.2.1). For the analysis of full-length S-binding IgG levels, all available IgG data for participants receiving frozen-liquid BNT162b2 in MDVs from Part 1 will be used. For the analysis of SARS-CoV-2 neutralizing titers, a random sample of approximately 30 age-matched participants receiving frozen-liquid BNT162b2 in MDVs will be selected from Part 1 of the study. |
| | GMCs of full-length S-binding IgG levels and/or GMTs of SARS-CoV-2 neutralizing titers |
| | For full-length S-binding IgG levels and/or SARS-CoV-2 neutralizing titers, GMCs/GMTs and 2-sided 95% CIs will be provided for each vaccine group in Part 2 of the study (frozen-liquid BNT162b2 with LNP size at the upper end of specification and RTU formulation) at baseline (before Dose 1) and at 1 month after Dose 2. |
| | Statistical methods are described in Section 9.4.1.2.2. |
| | GMFRs of full-length S-binding IgG levels and/or SARS-CoV-2 neutralizing titers |
| | For full-length S-binding IgG levels, the GMFRs and 2-sided 95% CIs will be provided for each vaccine group in Part 2 of the study (frozen-liquid BNT162b2 with LNP size at the upper end of specification and RTU formulation) from baseline (before Dose 1) to 1 month after Dose 2. |

| Endpoint | Statistical Analysis Methods |
|---|---|
| | GMFRs will be limited to participants with nonmissing values prior to the first dose and at the postvaccination time point. The statistical methods are described in Section 9.4.1.2.3. |
| | GMCs of full-length S-binding IgG levels and/or GMTs of SARS-CoV-2 neutralizing titers for participants receiving the third dose |
| | For full-length S-binding IgG levels and/or SARS-CoV-2 neutralizing titers, GMCs/GMTs and 2-sided 95% CIs will be provided for Dose 3 evaluable immunogenicity participants at baseline (before Dose 1), 1 month after Dose 2, prior to Dose 3, and 1 month after Dose 3. |
| | Statistical methods are described in Section 9.4.1.2.2. |
| | GMFRs of full-length S-binding IgG levels and/or SARS-CoV-2 neutralizing titers for participants receiving the third dose |
| | For full-length S-binding IgG levels and/or SARS-CoV-2 neutralizing titers, the GMFRs from prior to Dose 3 to 1 month after Dose 3 and 2-sided 95% CIs will be provided for participants receiving the third dose. |
| | GMFRs will be limited to participants with nonmissing values prior to Dose 3 and at 1 month after Dose 3. The statistical methods are described in Section 9.4.1.2.3. |

#### 9.5. Interim Analyses

No formal interim analysis will be conducted for this study. Statistical analyses will be carried out when the final data for specified objectives for a given study part are available while the study is ongoing.

## 9.6. Data Monitoring Committee or Other Independent Oversight Committee

This study will use a DMC. The DMC is independent of the study team and includes external members. The DMC charter describes the role of the DMC in more detail.

The DMC will be responsible for ongoing monitoring of the safety of participants in the study according to the charter. This may include, but is not limited to:

- Contemporaneous review of related AEs up to 1 month after completion of the vaccination schedule,
- Contemporaneous review of all SAEs up to 1 month after completion of the vaccination schedule.

The recommendations made by the DMC to alter the conduct of the study will be forwarded to the appropriate Pfizer personnel for final decision. Pfizer will forward such decisions, which may include summaries of aggregate analyses of safety data, to regulatory authorities, as appropriate.

#### 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

## 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations

## 10.1.1. Regulatory and Ethical Considerations

This study will be conducted in accordance with the protocol and with the following:

- Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and CIOMS International Ethical Guidelines;
- Applicable ICH GCP guidelines;
- Applicable laws and regulations, including applicable privacy laws.

The protocol, protocol amendments, ICD, SRSD(s), and other relevant documents (eg, advertisements) must be reviewed and approved by the sponsor and submitted to an IRB/EC by the investigator and reviewed and approved by the IRB/EC before the study is initiated.

Any amendments to the protocol will require IRB/EC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.

The investigator will be responsible for the following:

- Providing written summaries of the status of the study to the IRB/EC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC;
- Notifying the IRB/EC of SAEs or other significant safety findings as required by IRB/EC procedures;
- Providing oversight of the conduct of the study at the site and adherence to requirements of 21 CFR, ICH guidelines, the IRB/EC, European regulation 536/2014 for clinical studies (if applicable), and all other applicable local regulations.

## 10.1.1.1. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP

In the event of any prohibition or restriction imposed (ie, clinical hold) by an applicable regulatory authority in any area of the world, or if the investigator is aware of any new information that might influence the evaluation of the benefits and risks of the study intervention, Pfizer should be informed immediately.

In addition, the investigator will inform Pfizer immediately of any urgent safety measures taken by the investigator to protect the study participants against any immediate hazard, and of any serious breaches of this protocol or of ICH GCP that the investigator becomes aware of.

#### 10.1.2. Financial Disclosure

Investigators and subinvestigators will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### 10.1.3. Informed Consent Process

The investigator or his/her representative will explain the nature of the study to the participant and answer all questions regarding the study. The participant should be given sufficient time and opportunity to ask questions and to decide whether or not to participate in the trial.

Participants must be informed that their participation is voluntary. Participants will be required to sign a statement of informed consent that meets the requirements of 21 CFR 50, local regulations, ICH guidelines, HIPAA requirements, where applicable, and the IRB/EC or study center.

The investigator must ensure that each study participant is fully informed about the nature and objectives of the study, the sharing of data related to the study, and possible risks associated with participation, including the risks associated with the processing of the participant's personal data.

The participant must be informed that his/her personal study-related data will be used by the sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant.

The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB/EC members, and by inspectors from regulatory authorities.

The investigator further must ensure that each study participant is fully informed about his or her right to access and correct his or her personal data and to withdraw consent for the processing of his or her personal data.

The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICD.

Participants must be reconsented to the most current version of the ICD(s) during their participation in the study.

A copy of the ICD(s) must be provided to the participant. Participants who are rescreened are required to sign a new ICD.
Unless prohibited by local requirements or IRB/EC decision, the ICD will contain a separate section that addresses the use of samples for optional additional research. The optional additional research does not require the collection of any further samples. The investigator or authorized designee will explain to each participant the objectives of the additional research. Participants will be told that they are free to refuse to participate and may withdraw their consent at any time and for any reason during the storage period.

#### 10.1.4. Data Protection

All parties will comply with all applicable laws, including laws regarding the implementation of organizational and technical measures to ensure protection of participant data.

Participants' personal data will be stored at the study site in encrypted electronic and/or paper form and will be password protected or secured in a locked room to ensure that only authorized study staff have access. The study site will implement appropriate technical and organizational measures to ensure that the personal data can be recovered in the event of disaster. In the event of a potential personal data breach, the study site will be responsible for determining whether a personal data breach has in fact occurred and, if so, providing breach notifications as required by law.

To protect the rights and freedoms of participants with regard to the processing of personal data, participants will be assigned a single, participant-specific numerical code. Any participant records or data sets that are transferred to the sponsor will contain the numerical code; participant names will not be transferred. All other identifiable data transferred to the sponsor will be identified by this single, participant-specific code. The study site will maintain a confidential list of participants who participated in the study, linking each participant's numerical code to his or her actual identity and medical record identification. In case of data transfer, the sponsor will protect the confidentiality of participants' personal data consistent with the clinical study agreement and applicable privacy laws.

#### 10.1.5. Dissemination of Clinical Study Data

Pfizer fulfills its commitment to publicly disclose clinical study results through posting the results of studies on www.clinicaltrials.gov (ClinicalTrials.gov), the EudraCT, and/or www.pfizer.com, and other public registries in accordance with applicable local laws/regulations. In addition, Pfizer reports study results outside of the requirements of local laws/regulations pursuant to its SOPs.

In all cases, study results are reported by Pfizer in an objective, accurate, balanced, and complete manner and are reported regardless of the outcome of the study or the country in which the study was conducted.

#### www.clinicaltrials.gov

Pfizer posts clinical trial results on www.clinicaltrials.gov for Pfizer-sponsored interventional studies (conducted in patients) that evaluate the safety and/or efficacy of a product, regardless of the geographical location in which the study is conducted. These results are submitted for posting in accordance with the format and timelines set forth by US law.


#### EudraCT

Pfizer posts clinical trial results on EudraCT for Pfizer-sponsored interventional studies in accordance with the format and timelines set forth by EU requirements.

#### www.pfizer.com

Pfizer posts public disclosure synopses (CSR synopses in which any data that could be used to identify individual participants have been removed) on www.pfizer.com for Pfizer-sponsored interventional studies at the same time the corresponding study results are posted to www.clinicaltrials.gov.

#### Documents within marketing authorization packages/submissions

Pfizer complies with the European Union Policy 0070, the proactive publication of clinical data to the EMA website. Clinical data, under Phase 1 of this policy, includes clinical overviews, clinical summaries, CSRs, and appendices containing the protocol and protocol amendments, sample CRFs, and statistical methods. Clinical data, under Phase 2 of this policy, includes the publishing of individual participant data. Policy 0070 applies to new marketing authorization applications submitted via the centralized procedure since 01 January 2015 and applications for line extensions and for new indications submitted via the centralized procedure since 01 July 2015.

#### Data Sharing

Pfizer provides researchers secure access to patient-level data or full CSRs for the purposes of "bona-fide scientific research" that contributes to the scientific understanding of the disease, target, or compound class. Pfizer will make available data from these trials 24 months after study completion. Patient-level data will be anonymized in accordance with applicable privacy laws and regulations. CSRs will have personally identifiable information redacted.

Data requests are considered from qualified researchers with the appropriate competencies to perform the proposed analyses. Research teams must include a biostatistician. Data will not be provided to applicants with significant conflicts of interest, including individuals requesting access for commercial/competitive or legal purposes.

#### **10.1.6.** Data Quality Assurance

All participant data relating to the study will be recorded on printed or electronic CRF unless transmitted to the sponsor or designee electronically (eg, laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the CRF.

The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF.

The investigator must ensure that the CRFs are securely stored at the study site in encrypted electronic and/or paper form and are password protected or secured in a locked room to prevent access by unauthorized third parties.

The investigator must permit study-related monitoring, audits, IRB/EC review, and regulatory agency inspections and provide direct access to source data documents. This verification may also occur after study completion. It is important that the investigator(s) and their relevant personnel are available during the monitoring visits and possible audits or inspections and that sufficient time is devoted to the process.

Monitoring details describing strategy (eg, risk-based initiatives in operations and quality such as risk management and mitigation strategies and analytical risk-based monitoring), methods, responsibilities, and requirements, including handling of noncompliance issues and monitoring techniques (central, remote, or on-site monitoring), are provided in the monitoring plan.

The sponsor or designee is responsible for the data management of this study, including quality checking of the data.

Study monitors will perform ongoing source data verification to confirm that data entered into the CRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.

Records and documents, including signed ICDs, pertaining to the conduct of this study must be retained by the investigator for 15 years after study completion unless local regulations or institutional policies require a longer retention period. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor. The investigator must ensure that the records continue to be stored securely for as long as they are maintained.

When participant data are to be deleted, the investigator will ensure that all copies of such data are promptly and irrevocably deleted from all systems.

The investigator(s) will notify the sponsor or its agents immediately of any regulatory inspection notification in relation to the study. Furthermore, the investigator will cooperate with the sponsor or its agents to prepare the investigator site for the inspection and will allow the sponsor or its agent, whenever feasible, to be present during the inspection. The investigator site and investigator will promptly resolve any discrepancies that are identified between the study data and the participant's medical records. The investigator will promptly provide copies of the inspection findings to the sponsor or its agent. Before response submission to the regulatory authorities, the investigator will provide the sponsor or its agents with an opportunity to review and comment on responses to any such findings.

#### 10.1.7. Source Documents

Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator site.

Data reported on the CRF or entered in the eCRF that are from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.

Definition of what constitutes source data can be found in the study monitoring plan.

Description of the use of computerized system is documented in the data management plan.

#### 10.1.8. Study and Site Start and Closure

The study start date is the date on which the clinical study will be open for recruitment of participants.

The first act of recruitment is the date of the first participant's first visit and will be the study start date.

The sponsor designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time upon notification to the sponsor or designee if requested to do so by the responsible IRB/EC or if such termination is required to protect the health of study participants.

Reasons for the early closure of a study site by the sponsor may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/EC or local health authorities, the sponsor's procedures, or GCP guidelines;
- Inadequate recruitment of participants by the investigator;
- Discontinuation of further study intervention development.

If the study is prematurely terminated or suspended, the sponsor shall promptly inform the investigators, the ECs/IRBs, the regulatory authorities, and any CRO(s) used in the study of the reason for termination or suspension, as specified by the applicable regulatory requirements. The investigator shall promptly inform the participant and should assure appropriate participant therapy and/or follow-up.

Study termination is also provided for in the clinical study agreement. If there is any conflict between the contract and this protocol, the contract will control as to termination rights.

#### 10.1.9. Publication Policy

The results of this study may be published or presented at scientific meetings by the investigator after publication of the overall study results or 1 year after the end of the study (or study termination), whichever comes first.

The investigator agrees to refer to the primary publication in any subsequent publications such as secondary manuscripts, and submits all manuscripts or abstracts to the sponsor 30 days before submission. This allows the sponsor to protect proprietary information and to provide comments and the investigator will, on request, remove any previously undisclosed confidential information before disclosure, except for any study- or Pfizer intervention-related information necessary for the appropriate scientific presentation or understanding of the study results.

For all publications relating to the study, the investigator will comply with recognized ethical standards concerning publications and authorship, including those established by the International Committee of Medical Journal Editors.

The sponsor will comply with the requirements for publication of the overall study results covering all investigator sites. In accordance with standard editorial and ethical practice, the sponsor will support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement.

Authorship of publications for the overall study results will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

If publication is addressed in the clinical study agreement, the publication policy set out in this section will not apply.

#### 10.1.10. Sponsor's Qualified Medical Personnel

The contact information for the sponsor's appropriately qualified medical personnel for the study is documented in the study contact list located in the supporting study documentation or other electronic system.

To facilitate access to appropriately qualified medical personnel on study-related medical questions or problems, participants are provided with a contact card at the time of informed consent. The contact card contains, at a minimum, protocol and study intervention identifiers, participant numbers, contact information for the investigator site, and contact details for a contact center in the event that the investigator site staff cannot be reached to provide advice on a medical question or problem originating from another healthcare professional not involved in the participant's participation in the study. The contact number can also be used by investigator staff if they are seeking advice on medical questions or

problems; however, it should be used only in the event that the established communication pathways between the investigator site and the study team are not available. It is therefore intended to augment, but not replace, the established communication pathways between the investigator site and the study team for advice on medical questions or problems that may arise during the study. The contact number is not intended for use by the participant directly, and if a participant calls that number, he or she will be directed back to the investigator site.

#### 10.2. Appendix 2: Clinical Laboratory Tests

A pregnancy test will be performed at times defined in the SoA section of this protocol: Visit 1 (Vaccination 1/Day 1) and Visit 2 (Vaccination 2/19-23 days after Visit 1) as well as at Visit 101 for participants receiving Dose 3.

• Pregnancy test (β-hCG): Local urine testing will be standard for the protocol unless serum testing is required by local regulation or IRB/EC for female participants of childbearing potential.

Unscheduled clinical laboratory measurements may be obtained at any time during the study to assess any perceived safety issues. Investigators must document their review of each laboratory safety report.

## 10.3. Appendix 3: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### 10.3.1. Definition of AE

#### **AE Definition**

- An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.

#### **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (eg, ECG, radiological scans, vital sign measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator Any abnormal laboratory test results that meet any of the conditions below must be recorded as an AE:
  - Is associated with accompanying symptoms.
  - Requires additional diagnostic testing or medical/surgical intervention.
  - Leads to a change in study dosing (outside of any protocol-specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy.
- Exacerbation of a chronic or intermittent preexisting condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study intervention administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose per se will not be reported as an AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.

#### **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments which are associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of preexisting disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### 10.3.2. Definition of SAE

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met (eg, hospitalization for signs/symptoms of the disease under study, death due to progression of disease).

#### An SAE is defined as any untoward medical occurrence that, at any dose:

#### a. Results in death

#### b. Is life-threatening

The term "life-threatening" in the definition of "serious" refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it were more severe.

#### c. Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.

Hospitalization for elective treatment of a preexisting condition that did not worsen from baseline is not considered an AE.

#### d. Results in persistent disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (eg, sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### e. Is a congenital anomaly/birth defect

#### f. Other situations:

- Medical or scientific judgment should be exercised in deciding whether SAE
  reporting is appropriate in other situations such as important medical events that
  may not be immediately life-threatening or result in death or hospitalization but may
  jeopardize the participant or may require medical or surgical intervention to prevent
  one of the other outcomes listed in the above definition. These events should
  usually be considered serious.
- Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.
- Suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic, is considered serious. The event may be suspected from clinical symptoms or laboratory findings indicating an infection in a patient exposed to a Pfizer product. The terms "suspected transmission" and "transmission" are considered synonymous. These cases are considered unexpected and handled as serious expedited cases by pharmacovigilance personnel. Such cases are also considered for reporting as product defects, if appropriate.

#### 10.3.3. Recording/Reporting and Follow-up of AEs and/or SAEs

#### AE and SAE Recording/Reporting

The table below summarizes the requirements for recording adverse events on the CRF and for reporting serious adverse events on the Vaccine SAE Reporting Form to Pfizer Safety. These requirements are delineated for 3 types of events: (1) SAEs; (2) nonserious adverse events (AEs); and (3) exposure to the study intervention under study during pregnancy or breastfeeding, and occupational exposure.

It should be noted that the Vaccine SAE Reporting Form for reporting of SAE information is not the same as the AE page of the CRF. When the same data are collected, the forms must be completed in a consistent manner. AEs should be recorded using concise medical terminology and the same AE term should be used on both the CRF and the Vaccine SAE Reporting Form for reporting of SAE information.

| Safety Event | Recorded on the CRF | Reported on the Vaccine<br>SAE Reporting Form to<br>Pfizer Safety Within 24<br>Hours of Awareness |
|---|---|---|
| SAE | All | All |
| Nonserious AE | All | None |
| Exposure to the study intervention under study | All AEs/SAEs associated with exposure during | All (and EDP supplemental form for EDP) |
| during pregnancy or<br>breastfeeding, and<br>occupational exposure | pregnancy or breastfeeding | Note: Include all SAEs associated with exposure |
| | Occupational exposure is not recorded. | during pregnancy or<br>breastfeeding. Include all<br>AEs/SAEs associated with<br>occupational exposure. |

- When an AE/SAE occurs, it is the responsibility of the investigator to review all documentation (eg, hospital progress notes, laboratory reports, and diagnostic reports) related to the event.
- The investigator will then record all relevant AE/SAE information in the CRF.
- It is **not** acceptable for the investigator to send photocopies of the participant's medical records to Pfizer Safety in lieu of completion of the Vaccine SAE Reporting Form/AE/SAE CRF page.
- There may be instances when copies of medical records for certain cases are requested by Pfizer Safety. In this case, all participant identifiers, with the

exception of the participant number, will be redacted on the copies of the medical records before submission to Pfizer Safety.

• The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.

#### **Assessment of Intensity**

The investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to 1 of the following categories:

| GRADE | If required on the AE page of the CRF, the investigator will use the adjectives MILD, MODERATE, SEVERE, or LIFE-THREATENING to describe the maximum intensity of the AE. For purposes of consistency, these intensity grades are defined as follows: | |
|---|---|---|
| 1 | MILD | Does not interfere with participant's usual function. |
| 2 | MODERATE | Interferes to some extent with participant's usual function. |
| 3 | SEVERE | Interferes significantly with participant's usual function. |
| 4 | LIFE-THREATENING | Life-threatening consequences; urgent intervention indicated. |

#### **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE/SAE.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other
  risk factors, as well as the temporal relationship of the event to study intervention
  administration, will be considered and investigated.
- The investigator will also consult the IB and/or product information, for marketed products, in his/her assessment.
- For each AE/SAE, the investigator <u>must</u> document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to the sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.
- If the investigator does not know whether or not the study intervention caused the event, then the event will be handled as "related to study intervention" for reporting purposes, as defined by the sponsor. In addition, if the investigator determines that an SAE is associated with study procedures, the investigator must record this causal relationship in the source documents and CRF, and report such an assessment in the dedicated section of the Vaccine SAE Reporting Form and in accordance with the SAE reporting requirements.

#### Follow-up of AEs and SAEs

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by the sponsor to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other healthcare providers.
- If a participant dies during participation in the study or during a recognized follow-up period, the investigator will provide Pfizer Safety with a copy of any postmortem findings including histopathology.
- New or updated information will be recorded in the originally completed CRF.
- The investigator will submit any updated SAE data to the sponsor within 24 hours of receipt of the information.

#### 10.3.4. Reporting of SAEs

#### SAE Reporting to Pfizer Safety via Vaccine SAE Reporting Form

- Facsimile transmission of the Vaccine SAE Reporting Form is the preferred method to transmit this information to Pfizer Safety.
- In circumstances when the facsimile is not working, notification by telephone is acceptable with a copy of the Vaccine SAE Reporting Form sent by overnight mail or courier service.
- Initial notification via telephone does not replace the need for the investigator to complete and sign the Vaccine SAE Reporting Form pages within the designated reporting time frames.

#### 10.4. Appendix 4: Contraceptive Guidance

#### 10.4.1. Male Participant Reproductive Inclusion Criteria

Male participants are eligible to participate if they agree to the following requirements during the intervention period and for at least 28 days after the last dose of study intervention, which corresponds to the time needed to eliminate reproductive safety risk of the study intervention(s):

• Refrain from donating sperm.

#### PLUS either:

• Be abstinent from heterosexual intercourse with a female of childbearing potential as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.

#### OR

- Must agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person.
- In addition to male condom use, a highly effective method of contraception may be considered in WOCBP partners of male participants (refer to the list of highly effective methods below in Section 10.4.4).

#### 10.4.2. Female Participant Reproductive Inclusion Criteria

A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:

• Is not a WOCBP (see definitions below in Section 10.4.3).

#### OR

• Is a WOCBP and using an <u>acceptable</u> contraceptive method as described below during the intervention period (for a minimum of 28 days after the last dose of study intervention). The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

#### 10.4.3. Woman of Childbearing Potential

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

If fertility is unclear (eg, amenorrhea in adolescents or athletes) and a menstrual cycle cannot be confirmed before the first dose of study intervention, additional evaluation should be considered.

Women in the following categories are not considered WOCBP:

- 1. Premenopausal female with 1 of the following:
  - Documented hysterectomy;
  - Documented bilateral salpingectomy;
  - Documented bilateral oophorectomy.

For individuals with permanent infertility due to an alternate medical cause other than the above, (eg, mullerian agenesis, androgen insensitivity), investigator discretion should be applied to determining study entry.

Note: Documentation for any of the above categories can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview. The method of documentation should be recorded in the participant's medical record for the study.

#### 2. Postmenopausal female:

- A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. In addition, a
  - high FSH level in the postmenopausal range must be used to confirm a postmenopausal state in women under 60 years of age and not using hormonal contraception or HRT.
  - Female on HRT and whose menopausal status is in doubt will be required to use one of the nonestrogen hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

#### 10.4.4. Contraception Methods

Contraceptive use by men or women should be consistent with local availability/regulations regarding the use of contraceptive methods for those participating in clinical trials.

- 1. Implantable progestogen-only hormone contraception associated with inhibition of ovulation.
- 2. Intrauterine device.
- 3. Intrauterine hormone-releasing system.
- 4. Bilateral tubal occlusion.
- 5. Vasectomized partner:
  - Vasectomized partner is a highly effective contraceptive method provided that the
    partner is the sole sexual partner of the woman of childbearing potential and the
    absence of sperm has been confirmed. If not, an additional highly effective method
    of contraception should be used. The spermatogenesis cycle is approximately
    90 days.
- 6. Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation:
  - Oral:
  - Intravaginal;
  - Transdermal;
  - Injectable.
- 7. Progestogen-only hormone contraception associated with inhibition of ovulation:
  - Oral;
  - Injectable.
- 8. Sexual abstinence:
  - Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

- 9. Progestogen-only oral hormonal contraception where inhibition of ovulation is not the primary mode of action.
- 10. Male or female condom with or without spermicide.
- 11. Cervical cap, diaphragm, or sponge with spermicide.
- 12. A combination of male condom with either cervical cap, diaphragm, or sponge with spermicide (double-barrier methods).

# 10.5. Appendix 5: Liver Safety: Suggested Actions and Follow-up Assessments Potential Cases of Drug-Induced Liver Injury

Humans exposed to a drug who show no sign of liver injury (as determined by elevations in transaminases) are termed "tolerators," while those who show transient liver injury, but adapt are termed "adaptors." In some participants, transaminase elevations are a harbinger of a more serious potential outcome. These participants fail to adapt and therefore are "susceptible" to progressive and serious liver injury, commonly referred to as DILI. Participants who experience a transaminase elevation above 3 × ULN should be monitored more frequently to determine if they are an "adaptor" or are "susceptible."

LFTs are not required as a routine safety monitoring procedure in this study. However, should an investigator deem it necessary to assess LFTs because a participant presents with clinical signs/symptoms, such LFT results should be managed and followed as described below.

In the majority of DILI cases, elevations in AST and/or ALT precede TBili elevations (>2 × ULN) by several days or weeks. The increase in TBili typically occurs while AST/ALT is/are still elevated above 3 × ULN (ie, AST/ALT and TBili values will be elevated within the same laboratory sample). In rare instances, by the time TBili elevations are detected, AST/ALT values might have decreased. This occurrence is still regarded as a potential DILI. Therefore, abnormal elevations in either AST OR ALT in addition to TBili that meet the criteria outlined below are considered potential DILI (assessed per Hy's law criteria) cases and should always be considered important medical events, even before all other possible causes of liver injury have been excluded.

The threshold of laboratory abnormalities for a potential DILI case depends on the participant's individual baseline values and underlying conditions. Participants who present with the following laboratory abnormalities should be evaluated further as potential DILI (Hy's law) cases to definitively determine the etiology of the abnormal laboratory values:

- Participants with AST/ALT and TBili baseline values within the normal range who subsequently present with AST OR ALT values >3 × ULN AND a TBili value >2 × ULN with no evidence of hemolysis and an alkaline phosphatase value <2 × ULN or not available.
- For participants with baseline AST **OR** ALT **OR** TBili values above the ULN, the following threshold values are used in the definition mentioned above, as needed, depending on which values are above the ULN at baseline:
  - Preexisting AST or ALT baseline values above the normal range: AST or ALT values >2 times the baseline values AND >3 × ULN; or >8 × ULN (whichever is smaller).

• Preexisting values of TBili above the normal range: TBili level increased from baseline value by an amount of at least 1 × ULN **or** if the value reaches >3 × ULN (whichever is smaller).

Rises in AST/ALT and TBili separated by more than a few weeks should be assessed individually based on clinical judgment; any case where uncertainty remains as to whether it represents a potential Hy's law case should be reviewed with the sponsor.

The participant should return to the investigator site and be evaluated as soon as possible, preferably within 48 hours from awareness of the abnormal results. This evaluation should include laboratory tests, detailed history, and physical assessment.

In addition to repeating measurements of AST and ALT and TBili for suspected cases of Hy's law, additional laboratory tests should include albumin, CK, direct and indirect bilirubin, GGT, PT/INR, total bile acids, and alkaline phosphatase. Consideration should also be given to drawing a separate tube of clotted blood and an anticoagulated tube of blood for further testing, as needed, for further contemporaneous analyses at the time of the recognized initial abnormalities to determine etiology. A detailed history, including relevant information, such as review of ethanol, acetaminophen/paracetamol (either by itself or as a coformulated product in prescription or over-the-counter medications), recreational drug, supplement (herbal) use and consumption, family history, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and potential occupational exposure to chemicals, should be collected. Further testing for acute hepatitis A, B, C, D, and E infection and liver imaging (eg, biliary tract) and collection of serum samples for acetaminophen/paracetamol drug and/or protein adduct levels may be warranted.

All cases demonstrated on repeat testing as meeting the laboratory criteria of AST/ALT and TBili elevation defined above should be considered potential DILI (Hy's law) cases if no other reason for the LFT abnormalities has yet been found. Such potential DILI (Hy's law) cases are to be reported as SAEs, irrespective of availability of all the results of the investigations performed to determine etiology of the LFT abnormalities.

A potential DILI (Hy's law) case becomes a confirmed case only after all results of reasonable investigations have been received and have excluded an alternative etiology.

#### 10.6. Appendix 6: Abbreviations

The following is a list of abbreviations that may be used in the protocol.

| Abbreviation | Term |
|--------------|-------------------------------------------------------------|
| 2019-nCoV | novel coronavirus 2019 |
| AE | adverse event |
| AESI | adverse event of special interest |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| β-hCG | beta-human chorionic gonadotropin |
| CBER | Center for Biologics Evaluation and Research |
| CDC | Centers for Disease Control and Prevention |
| CFR | Code of Federal Regulations |
| CI | confidence interval |
| CIOMS | Council for International Organizations of Medical Sciences |
| CK | creatine kinase |
| CONSORT | Consolidated Standards of Reporting Trials |
| COVID-19 | coronavirus disease 2019 |
| CRF | case report form |
| CRO | contract research organization |
| CRU | clinical research unit |
| CSR | clinical study report |
| DILI | drug-induced liver injury |
| DMC | data monitoring committee |
| EC | ethics committee |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| e-diary | electronic diary |
| EDP | exposure during pregnancy |
| EMA | European Medicines Agency |
| EU | European Union |
| EUA | emergency use authorization |
| EudraCT | European Clinical Trials Database |
| FDA | Food and Drug Administration |
| FSH | follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GGT | gamma-glutamyl transferase |
| GMC | geometric mean concentration |
| GMFR | geometric mean fold rise |
| GMR | geometric mean ratio |
| GMT | geometric mean titer |
| HBV | hepatitis B virus |

| Abbreviation | Term |
|---|---|
| HCV | hepatitis C virus |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | human immunodeficiency virus |
| HRT | hormone replacement therapy |
| IB | investigator's brochure |
| ICD | informed consent document |
| ICH | International Council for Harmonisation |
| ID | identification |
| IgG | immunoglobulin G |
| IMP | investigational medicinal product |
| IND | investigational new drug |
| INR | international normalized ratio |
| IP manual | investigational product manual |
| IPAL | Investigational Product Accountability Log |
| IRB | institutional review board |
| IRT | interactive response technology |
| ISF | investigator site file |
| IWR | interactive Web-based response |
| JCVI | Joint Committee on Vaccination and Immunisation |
| LFT | liver function test |
| LLOQ | lower limit of quantitation |
| LNP | lipid nanoparticle |
| lyo | lyophilized |
| MDV | multidose vial |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MERS | Middle East respiratory syndrome |
| modRNA | nucleoside-modified messenger ribonucleic acid |
| N | SARS-CoV-2 nucleoprotein |
| N/A | not applicable |
| NAAT | nucleic acid amplification test |
| NIMP | noninvestigational medicinal product |
| P2 S | SARS-CoV-2 full-length, P2 mutant, prefusion spike glycoprotein |
| PI | principal investigator |
| PPE | personal protective equipment |
| PT | prothrombin time |
| PVC | premature ventricular contraction/complex |
| RCDC | reverse cumulative distribution curve |
| RNA | ribonucleic acid |
| RSV | respiratory syncytial virus |
| RT-PCR | reverse transcription-polymerase chain reaction |
| RTU | ready-to-use |

| Abbreviation | Term |
|--------------|-------------------------------------------------|
| S | spike protein |
| S1 | spike protein S1 subunit |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SARS | severe acute respiratory syndrome |
| SARS-CoV-2 | severe acute respiratory syndrome coronavirus 2 |
| SDV | single-dose vial |
| SSID | single subject identifier |
| SoA | schedule of activities |
| SOP | standard operating procedure |
| SRSD | single reference safety document |
| SUSAR | suspected unexpected serious adverse reaction |
| TBili | total bilirubin |
| Th 1 | T-helper type 1 |
| UK | United Kingdom |
| ULN | upper limit of normal |
| US | United States |
| VAED | vaccine-associated enhanced disease |
| WHO | World Health Organization |
| WOCBP | woman/women of childbearing potential |

#### 11. REFERENCES

- Virus Pathogen Resource (ViPR). Strain details for severe acute respiratory syndrome-related coronavirus strain Wuhan-Hu-1. Available from: https://www.viprbrc.org/brc/viprStrainDetails.spg?ncbiAccession=MN908947&decorat or=corona. Accessed: 11 Aug 2020.
- <sup>2</sup> Zhu N, Zhang D, Wang W, et al. A novel coronavirus from patients with pneumonia in China, 2019. N Engl J Med. 2020;382(8):727-33.
- World Health Organization. Timeline: WHO's COVID-19 response. Available from: https://www.who.int/emergencies/diseases/novel-coronavirus-2019/interactive-timeline#!. Accessed: 08 Jan 2021.
- World Health Organization. WHO Director-General's opening remarks at the media briefing on COVID-19. Available from: https://www.who.int/dg/speeches/detail/who-director-general-s-opening-remarks-at-the-media-briefing-on-covid-19---11-march-2020. Published: 11 Mar 2020. Accessed: 01 Apr 2020.
- COVID-19 dashboard by the Center for Systems Science and Engineering (CSSE) at Johns Hopkins University. Available from: https://gisanddata.maps.arcgis.com/apps/opsdashboard/index.html#/bda7594740fd40299 423467b48e9ecf6. Accessed: 08 Jan 2021.
- Rauch S, Jasny E, Schmidt KE, et al. New vaccine technologies to combat outbreak situations. Front Immunol. 2018;9:1963.
- Sahin U, Karikó K, Türeci Ö. mRNA-based therapeutics—developing a new class of drugs. Nat Rev Drug Discov. 2014;13(10):759-80.
- Polack FP, Thomas SJ, Kitchin N, et al. Safety and efficacy of the BNT162b2 mRNA Covid-19 vaccine. N Engl J Med. 2020;383(27):2603-15.
- Vaccines and Related Biological Products Advisory Committee. Vaccines and Related Biological Products Advisory Committee December 10, 2020, meeting: FDA Briefing Document Pfizer-BioNTech COVID-19 Vaccine. Silver Spring, MD: US Department of Health and Human Services, Food and Drug Administration; Dec 2020.
- Walsh EE, Frenck FW Jr, Falsey AR, et al. Safety and immunogenicity of two RNA-based Covid-19 vaccine candidates. N Engl J Med. 2020;383(25):2439-50. DOI: 10.1056/NEJMoa2027906.
- BioNTech RNA Pharmaceuticals GmbH. CorVAC/BNT162 investigator's brochure. Mainz, Germany: BioNTech RNA Pharmaceuticals GmbH; 12 Aug 2020.

- US Food and Drug Administration. Guidance for industry: toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials. Rockville, MD: Center for Biologics Evaluation and Research; Sep 2007.
- Centers for Disease Control and Prevention. Symptoms of coronavirus. Available from: https://www.cdc.gov/coronavirus/2019-ncov/symptoms-testing/symptoms.html. Updated: 13 May 2020. Accessed: 20 Oct 2020.

### **Document Approval Record**

| Document Name: | C4591020 Protocol Amendment 02 Clean Copy, 13 Sep 2021 |
|-----------------|--------------------------------------------------------|
| bootilion Hame. | C4591020 Protocol Amendment 02 Clean Copy, 13 Sep 2021 |

A PHASE 3, RANDOMIZED, OBSERVER-BLIND STUDY TO EVALU
ATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF MU
LTIPLE FORMULATIONS OF THE VACCINE CANDIDATE BNT162b2
AGAINST COVID 19 IN HEALTHY ADULTS 18 THROUGH 55 YEAR
S OF AGE

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|------------------------|
| PPD | 13-Sep-2021 12:41:34 | Business Line Approver |
| PPD | 13-Sep-2021 13:17:37 | Final Approval |